CLINICAL TRIAL: NCT01193335
Title: A Phase 4, Open-label Trial Describing The Safety, Tolerability, And Immunogenicity Of The 13 Valent Pneumococcal Conjugate Vaccine In Preterm Compared To Term Infants
Brief Title: Study Evaluating a 13-valent Pneumococcal Conjugate Vaccine in Preterm Compared to Term Infants.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B1851037; 6096A1-4001 (Other: Alias Study Number); 2009-017332-41 (EudraCT Number)
Record Dates: First submitted 2010-08-31; First posted 2010-09-01 (Estimated); Results first posted 2015-02-04 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2016-09

CONDITIONS: 13-valent Pneumococcal Vaccine; Premature Birth; Immunization; Safety
Keywords: 13-valent pneumococcal conjugate vaccine; premature; immunization; safety.
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: Preterm infants (Active Comparator): Infant born at < 37 weeks of gestation.
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine
- Group 2: Term infants (Active Comparator): Infants born at ≥ 37 weeks of gestation
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 13-valent pneumococcal conjugate vaccine — 13-valent pneumococcal conjugate vaccine will be administered at 2, 3, 4 and 12 months of age.
  Arms: Group 1: Preterm infants
Biological: 13-valent pneumococcal conjugate vaccine — 13-valent pneumococcal conjugate vaccine will be administered at 2, 3, 4 and 12 months of age.
  Arms: Group 2: Term infants

SUMMARY:
The purpose of this study is to describe the safety, tolerability, and immunogenicity of a 2,3,4 and 12 month schedule of the 13-valent pneumococcal conjugate vaccine when given to preterm infants with concomitant vaccines, compared to infants born at term.There will be a follow-up phase to assess the persistence of the antibody response at 24 and 36 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Infants between 42 and 98 days of age (approximately 2 months) at the time of enrollment.

Exclusion Criteria:

* Previous vaccination with pneumococcal vaccine,Haemophilus influenzae type B (Hib) conjugate vaccine, meningococcal type C conjugate vaccine, or diphtheria, tetanus, pertussis, or poliovirus vaccines.
* Previous anaphylactic reaction or allergy to any vaccine
* Contraindication to vaccination
* Known or suspected immune deficiency or immune suppression
* Major known congenital malformation or serious chronic disorder
* Significant neurological disorder
* Participation to another study

Ages: 42 Days to 98 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2010-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- Poland (6):
  - NZOZ "HIPOKRATES-II" Sp. z o.o., Krakow
  - Hanna Czajka Indywidualna Praktyka Specjalistyczna Lekarska, Krakow
  - SP ZOZ Wojewodzki Specjalistyczny Szpital im. W. Bieganskiego w Lodzi, Lodz
  - Specjalistyczny ZOZ nad Matka i Dzieckiem, Poznan
  - Szpital im. Sw. Jadwigi Slaskiej, Oddzial Pediatryczny, Trzebnica
  - Samodzielny Publiczny Szpital Kliniczny nr 1 we Wroclawiu, Wroclaw
- Spain (6):
  - Hospital Universitario de Santiago de Compostela, Santiago de Compostela, A Coruña
  - Complejo Hospitalario DE Torrecardenas, Almería, Almeria
  - Complexo Hospitalario Xeral Cies, Vigo, Pontevedra
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario de La Paz, Madrid
  - Complejo Hospitalario de Navarra, Pamplona

REFERENCES:
- [Derived] Martinon-Torres F, Wysocki J, Center KJ, Czajka H, Majda-Stanislawska E, Omenaca F, Concheiro-Guisan A, Gimenez-Sanchez F, Szenborn L, Blazquez-Gamero D, Moreno-Galarraga L, Giardina PC, Sun G, Gruber WC, Scott DA, Gurtman A. Circulating Antibody 1 and 2 Years After Vaccination With the 13-Valent Pneumococcal Conjugate Vaccine in Preterm Compared With Term Infants. Pediatr Infect Dis J. 2017 Mar;36(3):326-332. doi: 10.1097/INF.0000000000001428. PMID 27902652
- [Derived] Martinon-Torres F, Czajka H, Center KJ, Wysocki J, Majda-Stanislawska E, Omenaca F, Bernaola Iturbe E, Blazquez Gamero D, Concheiro-Guisan A, Gimenez-Sanchez F, Szenborn L, Giardina PC, Patterson S, Gruber WC, Scott DA, Gurtman A. 13-valent pneumococcal conjugate vaccine (PCV13) in preterm versus term infants. Pediatrics. 2015 Apr;135(4):e876-86. doi: 10.1542/peds.2014-2941. Epub 2015 Mar 16. PMID 25780077
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1851037&StudyName=Study%20Evaluating%20a%2013-valent%20Pneumococcal%20Conjugate%20Vaccine%20in%20Preterm%20Compared%20to%20Term%20Infants.

RESULTS

PARTICIPANT FLOW:
Groups:
- 13vPnC Group 1 (Preterm Infant): Preterm infant participants (gestational age [GA] less than [<] 37 weeks) received single 0.5 milliliter (mL) dose of 13-valent pneumococcal conjugate vaccine (13vPnC) intramuscularly at 2, 3, 4 months of age (infant series) and at 12 months of age (toddler dose). Preterm infant group was subdivided into Group 1A (GA greater than or equal to [>=] 32 weeks and <37 weeks), Group 1B (GA >=29 weeks and <32 weeks) and Group 1C (GA <29 weeks).
- 13vPnC Group 2 (Term Infant): Term infant participants (GA >=37 weeks) received single 0.5 mL dose of 13vPnC intramuscularly at 2, 3, 4 months of age (infant series) and at 12 months of age (toddler dose).
Period: Infant Series
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Started | 100 | 100
Completed | 100 | 100
Not Completed | 0 | 0
Period: After Infant Series
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Started | 100 | 100
Completed | 99 | 97
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — No Longer Met Eligibility Criteria | 0 | 1
Period: Toddler Dose
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Started | 99 | 97
Completed | 99 | 97
Not Completed | 0 | 0
Period: 1-Year Follow-up
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Started | 99 | 97
Completed | 88 | 88
Not Completed | 11 | 9
Not completed — No Longer Willing to Participate | 7 | 9
Not completed — Lost to Follow-up | 4 | 0
Period: 2-Year Follow-up
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Started | 88 | 88
Completed | 81 | 80
Not Completed | 7 | 8
Not completed — No Longer Willing to Participate | 5 | 6
Not completed — No Longer Met Eligibility Criteria | 2 | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis set included all participants who received at least 1 dose of 13vPnC.
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant) | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: months] | 1.8 (0.6) | 1.5 (0.5) | 1.7 (0.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 55 | 103
  Male | 52 | 45 | 97

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody Level Greater Than or Equal to (>=) 0.35 Microgram Per Milliliter (mcg/mL) 1 Month After Infant Series
Description: Percentage of participants achieving predefined antibody threshold >=0.35 mcg/mL along with the corresponding 95 percent (%) confidence interval (CI) for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) were presented. Exact 2-sided CI based on the observed proportion of participants. Here 'n' signifies participants with a determinate IgG concentration to the given serotype for each arm, respectively.
Time Frame: 1 month after the infant series
Population: Evaluable infant immunogenicity population included eligible participants who received all the assigned vaccinations (Infant Dose 1, 2 and 3), had blood drawn within required time frames, had at least 1 valid and determinate assay result for the proposed analysis, received no prohibited vaccines, and had no major protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Number analyzed (Participants) | 99 | 98
percentage of participants
  4 (n=99, 97) | 96.97 [91.40 to 99.37] | 98.97 [94.39 to 99.97]
  6B (n=99, 97) | 72.73 [62.85 to 81.20] | 87.63 [79.39 to 93.44]
  9V (n=99, 97) | 96.97 [91.40 to 99.37] | 96.91 [91.23 to 99.36]
  14 (n=99, 97) | 100.00 [96.34 to 100.00] | 97.94 [92.75 to 99.75]
  18C (n=99, 97) | 96.97 [91.40 to 99.37] | 94.85 [88.38 to 98.31]
  19F (n=99, 97) | 98.99 [94.50 to 99.97] | 98.97 [94.39 to 99.97]
  23F (n=99, 97 ) | 85.86 [77.41 to 92.05] | 92.78 [85.70 to 97.05]
  1 (n=99, 97) | 93.94 [87.27 to 97.74] | 95.88 [89.78 to 98.87]
  3 (n=99, 97) | 85.86 [77.41 to 92.05] | 90.72 [83.12 to 95.67]
  5 (n=99, 97) | 71.72 [61.78 to 80.31] | 90.72 [83.12 to 95.67]
  6A (n=98, 97) | 82.65 [73.69 to 89.56] | 94.85 [88.38 to 98.31]
  7F (n=99, 97) | 98.99 [94.50 to 99.97] | 98.97 [94.39 to 99.97]
  19A (n=99, 97) | 98.99 [94.50 to 99.97] | 98.97 [94.39 to 99.97]
Statistical Analysis 1: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 4: Exact 2-sided, 95% CI was computed based on the procedure of Chan and Zhang, using the standardized test statistics and gamma=0.000001; Test type: Superiority or Other; Percent difference = -2.00, 95% CI 2-sided [-7.65 to 2.88]
Statistical Analysis 2: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 6B: Exact 2-sided, 95% CI was computed based on the procedure of Chan and Zhang, using the standardized test statistics and gamma=0.000001; Test type: Superiority or Other; Percent difference = -14.90, 95% CI 2-sided [-26.40 to -3.21]
Statistical Analysis 3: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 9V: Exact 2-sided, 95% CI was computed based on the procedure of Chan and Zhang, using the standardized test statistics and gamma=0.000001; Test type: Superiority or Other; Percent difference = 0.06, 95% CI 2-sided [-5.84 to 6.05]
Statistical Analysis 4: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 14: Exact 2-sided, 95% CI was computed based on the procedure of Chan and Zhang, using the standardized test statistics and gamma=0.000001; Test type: Superiority or Other; Percent difference = 2.06, 95% CI 2-sided [-1.71 to 7.25]
Statistical Analysis 5: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 18C: Exact 2-sided, 95% CI was computed based on the procedure of Chan and Zhang, using the standardized test statistics and gamma=0.000001; Test type: Superiority or Other; Percent difference = 2.12, 95% CI 2-sided [-4.09 to 8.89]
Statistical Analysis 6: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 19F: Exact 2-sided, 95% CI was computed based on the procedure of Chan and Zhang, using the standardized test statistics and gamma=0.000001; Test type: Superiority or Other; Percent difference = 0.02, 95% CI 2-sided [-4.54 to 4.68]
Statistical Analysis 7: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 23F: Exact 2-sided, 95% CI was computed based on the procedure of Chan and Zhang, using the standardized test statistics and gamma=0.000001; Test type: Superiority or Other; Percent difference = -6.92, 95% CI 2-sided [-16.19 to 1.89]
Statistical Analysis 8: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 1: Exact 2-sided, 95% CI was computed based on the procedure of Chan and Zhang, using the standardized test statistics and gamma=0.000001; Test type: Superiority or Other; Percent difference = -1.94, 95% CI 2-sided [-9.07 to 4.86]
Statistical Analysis 9: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 3: Exact 2-sided, 95% CI was computed based on the procedure of Chan and Zhang, using the standardized test statistics and gamma=0.000001; Test type: Superiority or Other; Percent difference = -4.86, 95% CI 2-sided [-14.40 to 4.39]
Statistical Analysis 10: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 5: Exact 2-sided, 95% CI was computed based on the procedure of Chan and Zhang, using the standardized test statistics and gamma=0.000001; Test type: Superiority or Other; Percent difference = -19.00, 95% CI 2-sided [-30.10 to -7.16]
Statistical Analysis 11: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 6A: Exact 2-sided, 95% CI was computed based on the procedure of Chan and Zhang, using the standardized test statistics and gamma=0.000001; Test type: Superiority or Other; Percent difference = -12.19, 95% CI 2-sided [-21.66 to -3.26]
Statistical Analysis 12: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 7F: Exact 2-sided, 95% CI was computed based on the procedure of Chan and Zhang, using the standardized test statistics and gamma=0.000001; Test type: Superiority or Other; Percent difference = 0.02, 95% CI 2-sided [-4.54 to 4.68]
Statistical Analysis 13: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 19A: Exact 2-sided, 95% CI was computed based on the procedure of Chan and Zhang, using the standardized test statistics and gamma=0.000001; Test type: Superiority or Other; Percent difference = 0.02, 95% CI 2-sided [-4.54 to 4.68]

2. Primary Outcome: Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody 1 Month After the Infant Series
Description: Antibody geometric mean concentration (GMC) for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) were presented. GMC (13vPnC) and corresponding 2-sided 95% CIs were evaluated. GMCs were calculated using all participants with available data for the specified blood draw. CIs for GMC were back transformations of a CI based on the Student t distribution for the mean logarithm of the concentrations.
Time Frame: 1 month after the infant series
Population: Evaluable infant immunogenicity population. Here 'n' signifies participants with a determinate IgG concentration to the given serotype for each arm, respectively.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Number analyzed (Participants) | 99 | 98
mcg/mL
  4 (n=99, 97) | 1.96 [1.67 to 2.31] | 2.46 [2.04 to 2.97]
  6B (n=99, 97) | 0.73 [0.55 to 0.97] | 1.30 [1.00 to 1.67]
  9V (n=99, 97) | 1.26 [1.08 to 1.47] | 1.70 [1.45 to 2.00]
  14 (n=99, 97) | 7.48 [6.23 to 8.99] | 6.08 [4.82 to 7.67]
  18C (n=99, 97) | 1.93 [1.66 to 2.24] | 1.93 [1.62 to 2.29]
  19F (n=99, 97) | 2.21 [1.89 to 2.58] | 3.05 [2.62 to 3.55]
  23F (n=99, 97) | 0.86 [0.69 to 1.07] | 1.36 [1.10 to 1.68]
  1 (n=99, 97) | 1.26 [1.06 to 1.48] | 1.79 [1.50 to 2.13]
  3 (n=99, 97) | 0.83 [0.70 to 0.98] | 0.86 [0.75 to 1.00]
  5 (n=99, 97) | 0.56 [0.44 to 0.70] | 1.03 [0.87 to 1.22]
  6A (n=98, 97) | 1.22 [0.98 to 1.53] | 2.01 [1.65 to 2.46]
  7F (n=99, 97) | 2.14 [1.81 to 2.53] | 3.02 [2.63 to 3.48]
  19A (n=99, 97) | 2.85 [2.44 to 3.33] | 3.35 [2.85 to 3.94]
Statistical Analysis 1: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 4: Ratios of GMCs were calculated by back transforming the mean difference between vaccine groups on the logarithmic scale. CIs for the ratio were back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures; Test type: Superiority or Other; GMC ratio = 0.80, 95% CI 2-sided [0.62 to 1.02]
Statistical Analysis 2: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 6B: Ratios of GMCs were calculated by back transforming the mean difference between vaccine groups on the logarithmic scale. CIs for the ratio were back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures; Test type: Superiority or Other; GMC ratio = 0.56, 95% CI 2-sided [0.38 to 0.82]
Statistical Analysis 3: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 9V: Ratios of GMCs were calculated by back transforming the mean difference between vaccine groups on the logarithmic scale. CIs for the ratio were back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures; Test type: Superiority or Other; GMC ratio = 0.74, 95% CI 2-sided [0.59 to 0.93]
Statistical Analysis 4: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 14: Ratios of GMCs were calculated by back transforming the mean difference between vaccine groups on the logarithmic scale. CIs for the ratio were back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures; Test type: Superiority or Other; GMC ratio = 1.23, 95% CI 2-sided [0.92 to 1.65]
Statistical Analysis 5: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 18C: Ratios of GMCs were calculated by back transforming the mean difference between vaccine groups on the logarithmic scale. CIs for the ratio were back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures; Test type: Superiority or Other; GMC ratio = 1.00, 95% CI 2-sided [0.80 to 1.25]
Statistical Analysis 6: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 19F: Ratios of GMCs were calculated by back transforming the mean difference between vaccine groups on the logarithmic scale. CIs for the ratio were back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures; Test type: Superiority or Other; GMC ratio = 0.72, 95% CI 2-sided [0.58 to 0.90]
Statistical Analysis 7: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 23F: Ratios of GMCs were calculated by back transforming the mean difference between vaccine groups on the logarithmic scale. CIs for the ratio were back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures; Test type: Superiority or Other; GMC ratio = 0.64, 95% CI 2-sided [0.47 to 0.86]
Statistical Analysis 8: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 1: Ratios of GMCs were calculated by back transforming the mean difference between vaccine groups on the logarithmic scale. CIs for the ratio were back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures; Test type: Superiority or Other; GMC ratio = 0.70, 95% CI 2-sided [0.55 to 0.89]
Statistical Analysis 9: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 3: Ratios of GMCs were calculated by back transforming the mean difference between vaccine groups on the logarithmic scale. CIs for the ratio were back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures; Test type: Superiority or Other; GMC ratio = 0.96, 95% CI 2-sided [0.77 to 1.19]
Statistical Analysis 10: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 5: Ratios of GMCs were calculated by back transforming the mean difference between vaccine groups on the logarithmic scale. CIs for the ratio were back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures; Test type: Superiority or Other; GMC ratio = 0.54, 95% CI 2-sided [0.40 to 0.72]
Statistical Analysis 11: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 6A: Ratios of GMCs were calculated by back transforming the mean difference between vaccine groups on the logarithmic scale. CIs for the ratio were back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures; Test type: Superiority or Other; GMC ratio = 0.61, 95% CI 2-sided [0.45 to 0.82]
Statistical Analysis 12: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 7F: Ratios of GMCs were calculated by back transforming the mean difference between vaccine groups on the logarithmic scale. CIs for the ratio were back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures; Test type: Superiority or Other; GMC ratio = 0.71, 95% CI 2-sided [0.57 to 0.88]
Statistical Analysis 13: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 19: Ratios of GMCs were calculated by back transforming the mean difference between vaccine groups on the logarithmic scale. CIs for the ratio were back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures; Test type: Superiority or Other; GMC ratio = 0.85, 95% CI 2-sided [0.68 to 1.07]

3. Primary Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions Within 7 Days After Dose 1 Infant Series
Description: Local reactions were reported using an electronic diary. Tenderness was scaled as Any (tenderness present); Mild (hurts if gently touched with no crying); Moderate (hurts if gently touched with crying); Severe (causes limitation of limb movement). Redness and swelling were scaled as Any (redness or swelling present); Mild (0.5 centimeters [cm] to 2.0 cm); Moderate (2.5 to 7.0 cm); Severe (>7.0 cm). Participants may be represented in more than 1 category.
Time Frame: Within 7 days after Dose 1 of the infant series
Population: Safety population for Dose 1 infant series: all participants who received13vPnC Dose 1. Here 'N' (number of participants analyzed)=participants reporting yes for at least 1 day or no for all days for any local reaction.'n'=participants reporting yes for at least 1 day or no for all days for the specified local reaction for each group, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Number analyzed (Participants) | 98 | 92
percentage of participants
  Tenderness- Any (n=94, 88) | 48.9 | 42.0
  Tenderness- Mild (n=93, 88) | 46.2 | 31.8
  Tenderness- Moderate (n=90, 85) | 17.8 | 16.5
  Tenderness- Severe (n=86, 85) | 0.0 | 0.0
  Swelling- Any (n=94, 89) | 39.4 | 29.2
  Swelling- Mild (n=91, 89) | 37.4 | 28.1
  Swelling- Moderate (n=91, 85) | 8.8 | 8.2
  Swelling- Severe (n=86, 85) | 0.0 | 0.0
  Redness- Any (n=92, 87) | 33.7 | 29.9
  Redness- Mild (n=90, 87) | 32.2 | 28.7
  Redness- Moderate (n=88, 85) | 3.4 | 4.7
  Redness- Severe (n=86, 85) | 0.0 | 0.0

4. Primary Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions Within 7 Days After Dose 2 Infant Series
Description: as for outcome 3
Time Frame: Within 7 days after Dose 2 of the infant series
Population: Safety population for Dose 2 infant series: all participants who received 13vPnC Dose 2.Here 'N' (number of participants analyzed)=participants reporting yes for at least 1 day or no for all days for any local reaction.'n'=participants reporting yes for at least 1 day or no for all days for the specified local reaction for each group, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Number analyzed (Participants) | 89 | 89
percentage of participants
  Tenderness- Any (n=85, 88 ) | 48.2 | 38.6
  Tenderness- Mild (n=85, 84) | 43.5 | 31.0
  Tenderness- Moderate (n=77, 83) | 14.3 | 15.7
  Tenderness- Severe (n=73, 77) | 0.0 | 1.3
  Swelling- Any (n=84, 82) | 35.7 | 42.7
  Swelling- Mild (n=83, 82) | 33.7 | 42.7
  Swelling- Moderate (n=75, 76) | 8.0 | 2.6
  Swelling- Severe (n=73, 76) | 0.0 | 0.0
  Redness- Any (n=82, 82) | 28.0 | 40.2
  Redness- Mild (n=82, 82) | 28.0 | 37.8
  Redness- Moderate (n=73, 76) | 2.7 | 2.6
  Redness- Severe (n=73, 76) | 0.0 | 0.0

5. Primary Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions Within 7 Days After Dose 3 Infant Series
Description: as for outcome 3
Time Frame: Within 7 days after Dose 3 of the infant series
Population: Safety population for Dose 3 infant series: all participants who received 13vPnC Dose 3.Here 'N' (number of participants analyzed)=participants reporting yes for at least 1 day or no for all days for any local reaction.'n'=participants reporting yes for at least 1 day or no for all days for the specified local reaction for each group, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Number analyzed (Participants) | 87 | 90
percentage of participants
  Tenderness- Any (n=82, 84) | 39.0 | 28.6
  Tenderness- Mild (n=81, 84) | 35.8 | 26.2
  Tenderness- Moderate (n=75, 78) | 9.3 | 5.1
  Tenderness- Severe (n=73, 77) | 0.0 | 0.0
  Swelling- Any (n=83, 85) | 30.1 | 41.2
  Swelling- Mild (n=82, 85) | 26.8 | 41.2
  Swelling- Moderate (n=75, 79) | 5.3 | 5.1
  Swelling- Severe (n=73, 77) | 0.0 | 0.0
  Redness- Any (n=82, 87) | 32.9 | 46.0
  Redness- Mild (n=82, 87) | 32.9 | 46.0
  Redness- Moderate (n=74, 79) | 1.4 | 3.8
  Redness- Severe (n=73, 77) | 0.0 | 0.0

6. Primary Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions Within 7 Days After Toddler Dose
Description: as for outcome 3
Time Frame: Within 7 days after the toddler dose
Population: Safety population for Toddler Dose: all participants who received 13vPnC Toddler Dose. Here 'N' (number of participants analyzed)=participants reporting yes for at least 1 day or no for all days for any local reaction.'n'=participants reporting yes for at least 1 day or no for all days for the specified local reaction for each group, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Number analyzed (Participants) | 89 | 88
percentage of participants
  Tenderness- Any (n=86, 85) | 69.8 | 55.3
  Tenderness- Mild (n=86, 85) | 66.3 | 51.8
  Tenderness- Moderate (n=77, 70) | 20.8 | 11.4
  Tenderness- Severe (n=74, 69) | 2.7 | 0.0
  Swelling- Any (n=81, 80) | 43.2 | 35.0
  Swelling- Mild (n=80, 79) | 38.8 | 32.9
  Swelling- Moderate (n=76, 74) | 13.2 | 9.5
  Swelling- Severe (n=74, 69) | 1.4 | 0.0
  Redness- Any (n=85, 83) | 51.8 | 49.4
  Redness- Mild (n=85, 83) | 51.8 | 48.2
  Redness- Moderate (n=75, 75) | 6.7 | 10.7
  Redness- Severe (n=74, 69) | 0.0 | 0.0

7. Primary Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events Within 7 Days After Dose 1 Infant Series
Description: Systemic events (fever >=38 degrees Celsius [C], decreased appetite, increased sleep, and irritability or decreased sleep) and use of antipyretic medication were reported using an electronic diary. Decreased appetite was scaled as Any; Mild (loss of appetite but no decreased oral intake); Moderate (decreased oral intake); Severe (refusal to feed). Increased sleep was scaled as Any; Mild (increased or prolonged sleeping bouts); Moderate (slightly subdued interfering with daily activity); Severe (disabling not interested in usual daily activity). Irritability or decreased sleep was scaled as Any; Mild (easily consolable); Moderate (requiring increased attention); Severe (inconsolable; crying that cannot be comforted). Participants may be represented in more than 1 category.
Time Frame: Within 7 days after Dose 1 of the infant series
Population: Safety population for Dose 1 infant series: all participants who received 13vPnC Dose 1. Here 'N' (number of participants analyzed)=participants reporting yes for at least 1 day or no for all days for any event and 'n'=participants reporting yes for at least 1 day or no for all days for specified event for each group, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Number analyzed (Participants) | 98 | 99
percentage of participants
  Fever >=38 degrees C (n=86, 88) | 11.6 | 13.6
  Fever >=38 degrees C, =<39 degrees C (n=86, 88) | 10.5 | 13.6
  Fever >=39 degrees C, =<40 degrees C (n=86, 85) | 1.2 | 0.0
  Fever >40 degrees C (n=86, 85) | 0.0 | 0.0
  Decreased Appetite- Any (n=92, 89) | 60.9 | 41.6
  Decreased Appetite- Mild (n=91, 88) | 54.9 | 35.2
  Decreased Appetite- Moderate (n=88, 87) | 20.5 | 17.2
  Decreased Appetite- Severe (n=86, 85) | 1.2 | 0.0
  Increased Sleep- Any (n=96, 95) | 67.7 | 69.5
  Increased Sleep- Mild (n=96, 93) | 60.4 | 61.3
  Increased Sleep- Moderate (n=87, 88) | 29.9 | 30.7
  Increased Sleep- Severe (n=86, 85) | 2.3 | 2.4
  Irritability or Decreased Sleep- Any (n=95, 97) | 84.2 | 82.5
  Irritability or Decreased Sleep- Mild (n=93, 95) | 77.4 | 69.5
  Irritability or Decreased Sleep-Moderate (n=92, 91 | 43.5 | 47.3
  Irritability or Decreased Sleep- Severe (n=86, 85) | 8.1 | 5.9
  Use of Antipyretic Medication (n=90, 90) | 24.4 | 24.4

8. Primary Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events Within 7 Days After Dose 2 Infant Series
Description: as for outcome 7
Time Frame: Within 7 days after Dose 2 of the infant series
Population: Safety population for Dose 2 infant series: all participants who received 13vPnC Dose 2. Here 'N' (number of participants analyzed)=participants reporting yes for at least 1 day or no for all days for any event and 'n'=participants reporting yes for at least 1 day or no for all days for specified event for each group, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Number analyzed (Participants) | 97 | 96
percentage of participants
  Fever >=38 degrees C (n=79, 79) | 27.8 | 31.6
  Fever >=38 degrees C, =<39 degrees C (n=79, 79) | 27.8 | 30.4
  Fever >=39 degrees C, =<40 degrees C (n=73, 76) | 0.0 | 1.3
  Fever >40 degrees C (n=73, 76) | 0.0 | 0.0
  Decreased Appetite- Any (n=89, 84) | 61.8 | 46.4
  Decreased Appetite- Mild (n=88, 84) | 55.7 | 41.7
  Decreased Appetite- Moderate (n=79, 78) | 25.3 | 19.2
  Decreased Appetite- Severe (n=73, 76) | 1.4 | 0.0
  Increased Sleep- Any (n=85, 89 ) | 74.1 | 64.0
  Increased Sleep- Mild (n=83, 88) | 69.9 | 59.1
  Increased Sleep- Moderate (n=78, 78) | 34.6 | 29.5
  Increased Sleep- Severe (n=73, 76) | 2.7 | 1.3
  Irritability or Decreased Sleep- Any (n=95, 95) | 89.5 | 77.9
  Irritability or Decreased Sleep- Mild (n=90, 92) | 81.1 | 71.7
  Irritability or Decreased Sleep-Moderate (n=85, 86 | 64.7 | 44.2
  Irritability or Decreased Sleep- Severe (n=74, 76) | 17.6 | 2.6
  Use of Antipyretic Medication (n=84, 83) | 48.8 | 45.8

9. Primary Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events Within 7 Days After Dose 3 Infant Series
Description: as for outcome 7
Time Frame: Within 7 days after Dose 3 of the infant series
Population: Safety population for Dose 3 infant series: all participants who received 13vPnC Dose 3. Here 'N' (number of participants analyzed)=participants reporting yes for at least 1 day or no for all days for any event and 'n'=participants reporting yes for at least 1 day or no for all days for specified event for each group, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Number analyzed (Participants) | 94 | 95
percentage of participants
  Fever >=38 degrees C (n=79, 81) | 27.8 | 30.9
  Fever >=38 degrees C, =<39 degrees C (n=78, 81) | 26.9 | 30.9
  Fever >=39 degrees C, =<40 degrees C (n=75, 78) | 1.3 | 2.6
  Fever >40 degrees C (n=74, 77) | 0.0 | 0.0
  Decreased Appetite- Any (n=82, 84) | 48.8 | 47.6
  Decreased Appetite- Mild (n=82, 84) | 36.6 | 46.4
  Decreased Appetite- Moderate (n=74, 79) | 17.6 | 16.5
  Decreased Appetite- Severe (n=74, 77) | 1.4 | 1.3
  Increased Sleep- Any (n=88, 88 ) | 52.3 | 58.0
  Increased Sleep- Mild (n=88, 87) | 48.9 | 51.7
  Increased Sleep- Moderate (n=77, 80) | 16.9 | 20.0
  Increased Sleep- Severe (n=73, 77) | 1.4 | 1.3
  Irritability or Decreased Sleep- Any (n=92, 95) | 79.3 | 81.1
  Irritability or Decreased Sleep- Mild (n=90, 91) | 72.2 | 74.7
  Irritability or Decreased Sleep-Moderate (n=80,87) | 33.8 | 35.6
  Irritability or Decreased Sleep- Severe (n=74, 78) | 6.8 | 6.4
  Use of Antipyretic Medication (n=84, 81) | 40.5 | 38.3

10. Primary Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events Within 7 Days After Toddler Dose
Description: as for outcome 7
Time Frame: Within 7 days after the toddler dose
Population: Safety population for Toddler Dose: all participants who received 13vPnC Toddler Dose. Here 'N' (number of participants analyzed)=participants reporting yes for at least 1 day or no for all days for any event and 'n'=participants reporting yes for at least 1 day or no for all days for specified event for each group, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Number analyzed (Participants) | 93 | 92
percentage of participants
  Fever >=38 degrees C (n= 80, 78) | 28.8 | 43.6
  Fever >=38 degrees C, =<39 degrees C (n=80, 77) | 27.5 | 42.9
  Fever >=39 degrees C, =<40 degrees C (n=74, 71) | 1.4 | 4.2
  Fever >40 degrees C (n=74, 70) | 0.0 | 1.4
  Decreased Appetite- Any (n=87, 86) | 57.5 | 60.5
  Decreased Appetite- Mild (n=86, 84) | 50.0 | 56.0
  Decreased Appetite- Moderate (n=78, 73) | 25.6 | 23.3
  Decreased Appetite- Severe (n=75, 69) | 1.3 | 1.4
  Increased Sleep- Any (n=83, 86 ) | 57.8 | 65.1
  Increased Sleep- Mild (n=82, 84) | 53.7 | 59.5
  Increased Sleep- Moderate (n=76, 74) | 18.4 | 24.3
  Increased Sleep- Severe (n=74, 70) | 0.0 | 2.9
  Irritability or Decreased Sleep- Any (n=90, 91) | 84.4 | 80.2
  Irritability or Decreased Sleep- Mild (n=90, 89) | 74.4 | 76.4
  Irritability or Decreased Sleep-Moderate (n=78,80) | 44.9 | 45.0
  Irritability or Decreased Sleep- Severe (n=76, 69) | 6.6 | 4.3
  Use of Antipyretic Medication (n=82, 79) | 48.8 | 50.6

11. Primary Outcome: Percentage of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs): Infant Series
Description: An AE was any untoward medical occurrence in a participant who received vaccine without regard to possibility of causal relationship. SAE: an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial/prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Dose 1 up to 1 month after Dose 3 (infant series)
Population: Safety population for infant series included all participants who received at least 1 dose of 13vPnC during infant series.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Number analyzed (Participants) | 100 | 100
percentage of participants
  AEs | 59.0 | 55.0
  SAEs | 14.0 | 5.0
Statistical Analysis 1: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); AEs: Two sided Fisher exact test, was used to calculate difference between vaccine groups; Test type: Superiority or Other; p = 0.668, Fisher Exact
Statistical Analysis 2: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); SAEs: Two sided Fisher exact test, was used to calculate difference between vaccine groups; Test type: Superiority or Other; p = 0.051, Fisher Exact

12. Primary Outcome: Percentage of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs): After Infant Series
Description: as for outcome 11
Time Frame: 1 Month after Dose 3 of the infant series up to toddler dose
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Number analyzed (Participants) | 100 | 100
percentage of participants
  AEs | 18.0 | 15.0
  SAEs | 8.0 | 9.0
Statistical Analysis 1: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); AEs: Two sided Fisher exact test, was used to calculate difference between vaccine groups; Test type: Superiority or Other; p = 0.704, Fisher Exact
Statistical Analysis 2: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); SAEs: Two sided Fisher exact test, was used to calculate difference between vaccine groups; Test type: Superiority or Other; p > 0.99, Fisher Exact

13. Primary Outcome: Percentage of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs): Toddler Dose
Description: as for outcome 11
Time Frame: Toddler dose up to 1 Month after toddler dose
Population: Safety population for toddler dose included all participants who received 13vPnC toddler dose.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Number analyzed (Participants) | 99 | 97
percentage of participants
  AEs | 31.3 | 26.8
  SAEs | 2.0 | 1.0
Statistical Analysis 1: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); AEs: Two sided Fisher exact test, was used to calculate difference between vaccine groups; Test type: Superiority or Other; p = 0.531, Fisher Exact
Statistical Analysis 2: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); SAEs: Two sided Fisher exact test, was used to calculate difference between vaccine groups; Test type: Superiority or Other; p > 0.99, Fisher Exact

14. Primary Outcome: Percentage of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs): 1-Year Follow-up After Toddler Dose
Description: as for outcome 11
Time Frame: 1 month after toddler dose up to 1-year follow-up
Population: Safety population for 1-year follow-up after toddler dose included all participants who received 13vPnC toddler dose and had safety data available during specified follow-up period.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Number analyzed (Participants) | 99 | 97
percentage of participants
  AEs | 15.2 | 8.2
  SAEs | 13.1 | 8.2
Statistical Analysis 1: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); AEs: Two sided Fisher exact test, was used to calculate difference between vaccine groups; Test type: Superiority or Other; p = 0.183, Fisher Exact
Statistical Analysis 2: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); SAEs: Two sided Fisher exact test, was used to calculate difference between vaccine groups; Test type: Superiority or Other; p = 0.357, Fisher Exact

15. Primary Outcome: Percentage of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs): 2-Year Follow-up After Toddler Dose
Description: as for outcome 11
Time Frame: 1-year follow-up after toddler dose to 2-year follow-up after toddler dose
Population: Safety population for 2-year follow-up after toddler dose included all participants who received 13vPnC toddler dose and had safety data available during specified follow-up period.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Number analyzed (Participants) | 88 | 88
percentage of participants
  AEs | 8.0 | 10.2
  SAEs | 6.8 | 9.1
Statistical Analysis 1: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); AEs: Two sided Fisher exact test, was used to calculate difference between vaccine groups; Test type: Superiority or Other; p = 0.794, Fisher Exact
Statistical Analysis 2: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); SAEs: Two sided Fisher exact test, was used to calculate difference between vaccine groups; Test type: Superiority or Other; p = 0.782, Fisher Exact

16. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody From Toddler Pre-Dose to 1 Month After Toddler Dose
Description: GMFR for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) from before 13vPnC toddler dose to 1 month after 13vPnC toddler dose were computed using the logarithmically transformed assay results. CIs for GMFR were back transformations of confidence levels based on the Student t distribution for the mean logarithm of the fold rises. GMFRs were calculated using all participants with available data from both before 13vPnC toddler dose and after 13vPnC toddler dose blood draws.
Time Frame: Before 13vPnC Toddler Dose (pre-vaccination), 1 month after 13vPnC Toddler Dose
Population: Evaluable Toddler Immunogenicity Population. Here 'n' signifies participants with a determinate IgG antibody concentration to the given serotype for each arm, respectively.
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Groups:
- 13vPnC Group 1 (Preterm Infant): Preterm infant participants (GA <37 weeks) received single 0.5 mL dose of 13vPnC intramuscularly at 2, 3, 4 months of age (infant series) and at 12 months of age (toddler dose). Preterm infant group was subdivided into Group 1A (GA >=32 weeks and <37 weeks), Group 1B (GA >=29 weeks and <32 weeks) and Group 1C (GA <29 weeks).
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Number analyzed (Participants) | 88 | 88
fold rise
  4 (n= 83, 85) | 8.14 [6.61 to 10.04] | 9.61 [7.77 to 11.88]
  6B (n=80, 85) | 9.46 [7.81 to 11.45] | 7.61 [6.31 to 9.18]
  9V (n=83, 85) | 5.85 [5.05 to 6.78] | 4.92 [4.22 to 5.74]
  14 (n=83, 85) | 4.50 [3.76 to 5.38] | 4.65 [3.82 to 5.65]
  18C (n=83, 85) | 7.36 [6.29 to 8.61] | 9.14 [7.61 to 10.98]
  19F (n=83, 85) | 10.82 [8.88 to 13.17] | 12.31 [9.77 to 15.51]
  23F (n=79, 83) | 10.11 [8.13 to 12.57] | 10.15 [8.32 to 12.39]
  1 (n=83, 85) | 8.41 [6.94 to 10.20] | 9.98 [8.18 to 12.17]
  3 (n=81, 84) | 7.61 [5.79 to 10.01] | 5.23 [4.22 to 6.49]
  5 (n=80, 85) | 3.47 [3.04 to 3.97] | 3.46 [2.93 to 4.09]
  6A (n=83, 85) | 10.52 [8.75 to 12.64] | 7.72 [6.18 to 9.65]
  7F (n=83, 85) | 5.81 [5.12 to 6.61] | 6.07 [5.16 to 7.13]
  19A (n=83, 85) | 6.45 [5.39 to 7.72] | 5.59 [4.53 to 6.90]
Statistical Analysis 1: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 4: GMFR ratio was calculated by back transforming the GMFR difference between the groups on the logarithmic scale. CIs for the ratio were back transformations of a CI based on Student t distribution for the ratio difference of logarithms of the measures (Group 1 - Group 2); Test type: Superiority or Other; GMFR Ratio = 0.85, 95% CI 2-sided [0.63 to 1.14]
Statistical Analysis 2: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 6B: GMFR ratio was calculated by back transforming the GMFR difference between the groups on the logarithmic scale. CIs for the ratio were back transformations of a CI based on Student t distribution for the ratio difference of logarithms of the measures (Group 1 - Group 2); Test type: Superiority or Other; GMFR ratio = 1.24, 95% CI 2-sided [0.95 to 1.62]
Statistical Analysis 3: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 9V: GMFR ratio was calculated by back transforming the GMFR difference between the groups on the logarithmic scale. CIs for the ratio were back transformations of a CI based on Student t distribution for the ratio difference of logarithms of the measures (Group 1 - Group 2); Test type: Superiority or Other; GMFR ratio = 1.19, 95% CI 2-sided [0.96 to 1.47]
Statistical Analysis 4: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 14: GMFR ratio was calculated by back transforming the GMFR difference between the groups on the logarithmic scale. CIs for the ratio were back transformations of a CI based on Student t distribution for the ratio difference of logarithms of the measures (Group 1 - Group 2); Test type: Superiority or Other; GMFR ratio = 0.97, 95% CI 2-sided [0.74 to 1.26]
Statistical Analysis 5: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 18C: GMFR ratio was calculated by back transforming the GMFR difference between the groups on the logarithmic scale. CIs for the ratio were back transformations of a CI based on Student t distribution for the ratio difference of logarithms of the measures (Group 1 - Group 2); Test type: Superiority or Other; GMFR ratio = 0.80, 95% CI 2-sided [0.63 to 1.02]
Statistical Analysis 6: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 19F: GMFR ratio was calculated by back transforming the GMFR difference between the groups on the logarithmic scale. CIs for the ratio were back transformations of a CI based on Student t distribution for the ratio difference of logarithms of the measures (Group 1 - Group 2); Test type: Superiority or Other; GMFR ratio = 0.88, 95% CI 2-sided [0.65 to 1.19]
Statistical Analysis 7: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 23F: GMFR ratio was calculated by back transforming the GMFR difference between the groups on the logarithmic scale; Test type: Superiority or Other; GMFR ratio = 1.00, 95% CI 2-sided [0.74 to 1.33]
Statistical Analysis 8: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 1: GMFR ratio was calculated by back transforming the GMFR difference between the groups on the logarithmic scale; Test type: Superiority or Other; GMFR ratio = 0.84, 95% CI 2-sided [0.64 to 1.11]
Statistical Analysis 9: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 3: GMFR ratio was calculated by back transforming the GMFR difference between the groups on the logarithmic scale. CIs for the ratio were back transformations of a CI based on Student t distribution for the ratio difference of logarithms of the measures (Group 1 - Group 2); Test type: Superiority or Other; GMFR ratio = 1.46, 95% CI 2-sided [1.03 to 2.05]
Statistical Analysis 10: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 5: GMFR ratio was calculated by back transforming the GMFR difference between the groups on the logarithmic scale. CIs for the ratio were back transformations of a CI based on Student t distribution for the ratio difference of logarithms of the measures (Group 1 - Group 2); Test type: Superiority or Other; GMFR ratio = 1.00, 95% CI 2-sided [0.81 to 1.24]
Statistical Analysis 11: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 6A: GMFR ratio was calculated by back transforming the GMFR difference between the groups on the logarithmic scale. CIs for the ratio were back transformations of a CI based on Student t distribution for the ratio difference of logarithms of the measures (Group 1 - Group 2); Test type: Superiority or Other; GMFR ratio = 1.36, 95% CI 2-sided [1.02 to 1.82]
Statistical Analysis 12: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 7F: GMFR ratio was calculated by back transforming the GMFR difference between the groups on the logarithmic scale. CIs for the ratio were back transformations of a CI based on Student t distribution for the ratio difference of logarithms of the measures (Group 1 - Group 2); Test type: Superiority or Other; GMFR ratio = 0.96, 95% CI 2-sided [0.78 to 1.18]
Statistical Analysis 13: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 19A: GMFR ratio was calculated by back transforming the GMFR difference between the groups on the logarithmic scale. CIs for the ratio were back transformations of a CI based on Student t distribution for the ratio difference of logarithms of the measures (Group 1 - Group 2); Test type: Superiority or Other; GMFR ratio = 1.15, 95% CI 2-sided [0.88 to 1.52]

17. Secondary Outcome: Percentage of Participants Achieving Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody Level >=0.35 mcg/mL 1 Month After Infant Series: Group 1A, 1B, 1C
Description: Percentage of participants achieving predefined antibody threshold >=0.35 mcg/mL along with the corresponding 95 % CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) were presented. Exact 2-sided CI based on the observed proportion of participants. Here 'n' signifies participants with a determinate IgG concentration to the given serotype for each arm, respectively.
Time Frame: 1 Month After Infant Series
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 13vPnC Group 1A: Preterm infant participants with GA >=32 weeks and <37 weeks received single 0.5 mL dose of 13vPnC intramuscularly at 2, 3, 4 months of age (infant series) and at 12 months of age (toddler dose).
- 13vPnC Group 1B: Preterm infant participants with GA >=29 weeks and <32 weeks received single 0.5 mL dose of 13vPnC intramuscularly at 2, 3, 4 months of age (infant series) and at 12 months of age (toddler dose).
- 13vPnC Group 1C: Preterm participants with GA <29 weeks received single 0.5 mL dose of 13vPnC intramuscularly at 2, 3, 4 months of age (infant series) and at 12 months of age (toddler dose).
Arm/Group | 13vPnC Group 1A | 13vPnC Group 1B | 13vPnC Group 1C
Number analyzed (Participants) | 24 | 50 | 25
percentage of participants
  4 (n=24, 50, 25) | 100.00 [85.75 to 100.00] | 96.00 [86.29 to 99.51] | 96.00 [79.65 to 99.90]
  6B (n=24, 50, 25) | 79.17 [57.85 to 92.87] | 72.00 [57.51 to 83.77] | 68.00 [46.50 to 85.05]
  9V (n=24, 50, 25) | 95.83 [78.88 to 99.89] | 98.00 [89.35 to 99.95] | 96.00 [79.65 to 99.90]
  14 (n=24, 50, 25) | 100.00 [85.75 to 100.00] | 100.00 [92.89 to 100.00] | 100.00 [86.28 to 100.00]
  18C (n=24, 50, 25) | 100.00 [85.75 to 100.00] | 94.00 [83.45 to 98.75] | 100.00 [86.28 to 100.00]
  19F (n=24, 50, 25) | 100.00 [85.75 to 100.00] | 98.00 [89.35 to 99.95] | 100.00 [86.28 to 100.00]
  23F (n=24, 50, 25) | 91.67 [73.00 to 98.97] | 80.00 [66.28 to 89.97] | 92.00 [73.97 to 99.02]
  1 (n=24, 50, 25) | 100.00 [85.75 to 100.00] | 92.00 [80.77 to 97.78] | 92.00 [73.97 to 99.02]
  3 (n=24, 50, 25) | 87.50 [67.64 to 97.34] | 86.00 [73.26 to 94.18] | 84.00 [63.92 to 95.46]
  5 (n=24, 50, 25) | 79.17 [57.85 to 92.87] | 66.00 [51.23 to 78.79] | 76.00 [54.87 to 90.64]
  6A (n=24, 49, 25) | 95.83 [78.88 to 99.89] | 81.63 [67.98 to 91.24] | 72.00 [50.61 to 87.93]
  7F (n=24, 50, 25) | 100.00 [85.75 to 100.00] | 98.00 [89.35 to 99.95] | 100.00 [86.28 to 100.00]
  19A (n=24, 50, 25) | 100.00 [85.75 to 100.00] | 98.00 [89.35 to 99.95] | 100.00 [86.28 to 100.00]

18. Secondary Outcome: Percentage of Participants Achieving Serotype-specific Pneumococcal IgG Antibody Level ≥0.35 mcg/mL 1 Month After the Toddler Dose
Description: Percentage of participants achieving predefined antibody threshold >=0.35 mcg/mL along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) were presented. Exact 2-sided CI based on the observed proportion of participants. Here 'n' signifies participants with a determinate IgG antibody concentration to the given serotype for each arm, respectively.
Time Frame: 1 month after the toddler dose
Population: Evaluable Toddler Immunogenicity Population included eligible participants who received all the assigned vaccinations (Infant Dose 1, 2, 3 and toddler dose), had blood drawn within required time frames, had at least 1 valid and determinate assay result for the proposed analysis, received no prohibited vaccines, and had no major protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Number analyzed (Participants) | 88 | 88
percentage of participants
  4 (n= 86, 87) | 100.00 [95.80 to 100.00] | 100.00 [95.85 to 100.00]
  6B (n=86, 87) | 97.67 [91.85 to 99.72] | 100.00 [95.85 to 100.00]
  9V (n=86, 87) | 100.00 [95.80 to 100.00] | 100.00 [95.85 to 100.00]
  14 (n=86, 87) | 100.00 [95.80 to 100.00] | 100.00 [95.85 to 100.00]
  18C (n=86, 87) | 100.00 [95.80 to 100.00] | 98.85 [93.76 to 99.97]
  19F (n=86, 87) | 100.00 [95.80 to 100.00] | 100.00 [95.85 to 100.00]
  23F (n=86, 87) | 98.84 [93.69 to 99.97] | 100.00 [95.85 to 100.00]
  1 (n=86, 87) | 100.00 [95.80 to 100.00] | 100.00 [95.85 to 100.00]
  3 (n=85, 87) | 70.59 [59.71 to 79.98] | 79.31 [69.29 to 87.25]
  5 (n=86, 87) | 100.00 [95.80 to 100.00] | 100.00 [95.85 to 100.00]
  6A (n=86, 87) | 100.00 [95.80 to 100.00] | 100.00 [95.85 to 100.00]
  7F (n=86, 87) | 100.00 [95.80 to 100.00] | 100.00 [95.85 to 100.00]
  19A (n=86, 87) | 100.00 [95.80 to 100.00] | 100.00 [95.85 to 100.00]
Statistical Analysis 1: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Percent difference = 0.00, 95% CI 2-sided [-4.25 to 4.31]
Statistical Analysis 2: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Percent difference = -2.33, 95% CI 2-sided [-8.15 to 1.96]
Statistical Analysis 3: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; Percent difference = 0.00, 95% CI 2-sided [-4.25 to 4.31]
Statistical Analysis 4: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; Percent difference = 0.00, 95% CI 2-sided [-4.25 to 4.31]
Statistical Analysis 5: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; Percent difference = 1.15, 95% CI 2-sided [-3.13 to 6.24]
Statistical Analysis 6: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 1, analysis 6]; Test type: Superiority or Other; Percent difference = 0.00, 95% CI 2-sided [-4.25 to 4.31]
Statistical Analysis 7: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 1, analysis 7]; Test type: Superiority or Other; Percent difference = -1.16, 95% CI 2-sided [-6.32 to 3.10]
Statistical Analysis 8: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; Percent difference = 0.00, 95% CI 2-sided [-4.25 to 4.31]
Statistical Analysis 9: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; Percent difference = -8.72, 95% CI 2-sided [-21.93 to 4.42]
Statistical Analysis 10: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 1, analysis 10]; Test type: Superiority or Other; Percent difference = 0.00, 95% CI 2-sided [-4.25 to 4.31]
Statistical Analysis 11: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 1, analysis 11]; Test type: Superiority or Other; Percent difference = 0.00, 95% CI 2-sided [-4.25 to 4.31]
Statistical Analysis 12: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; Percent difference = 0.00, 95% CI 2-sided [-4.25 to 4.31]
Statistical Analysis 13: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 1, analysis 13]; Test type: Superiority or Other; Percent difference = 0.00, 95% CI 2-sided [-4.25 to 4.31]

19. Secondary Outcome: Percentage of Participants Achieving Serotype-specific Pneumococcal IgG Antibody Level >=0.35 mcg/mL 1 Month After Toddler Dose: Group 1A, 1B, 1C
Description: Percentage of participants achieving predefined antibody threshold >=0.35 mcg/mL along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) were presented. Exact 2-sided CI based on the observed proportion of participants.
Time Frame: 1 month after the toddler dose
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 13vPnC (Group 1A): Preterm infant participants with GA >=32 weeks and <37 weeks received single 0.5 mL dose of 13vPnC intramuscularly at 2, 3, 4 months of age (infant series) and at 12 months of age (toddler dose).
- 13vPnC (Group 1B): Preterm infant participants with GA >=29 weeks and <32 weeks received single 0.5 mL dose of 13vPnC intramuscularly at 2, 3, 4 months of age (infant series) and at 12 months of age (toddler dose).
- 13vPnC (Group 1C): Preterm infant participants with GA <29 weeks received single 0.5 mL dose of 13vPnC intramuscularly at 2, 3, 4 months of age (infant series) and at 12 months of age (toddler dose).
Arm/Group | 13vPnC (Group 1A) | 13vPnC (Group 1B) | 13vPnC (Group 1C)
Number analyzed (Participants) | 21 | 46 | 21
percentage of participants
  4 (n=21, 45, 20) | 100.00 [83.89 to 100.00] | 100.00 [92.13 to 100.00] | 100.00 [83.16 to 100.00]
  6B (n=21, 45, 20) | 100.00 [83.89 to 100.00] | 95.56 [84.85 to 99.46] | 100.00 [83.16 to 100.00]
  9V (n=21, 45, 20) | 100.00 [83.89 to 100.00] | 100.00 [92.13 to 100.00] | 100.00 [83.16 to 100.00]
  14 (n=21, 45, 20) | 100.00 [83.89 to 100.00] | 100.00 [92.13 to 100.00] | 100.00 [83.16 to 100.00]
  18C (n=21, 45, 20) | 100.00 [83.89 to 100.00] | 100.00 [92.13 to 100.00] | 100.00 [83.16 to 100.00]
  19F (n=21, 45, 20) | 100.00 [83.89 to 100.00] | 100.00 [92.13 to 100.00] | 100.00 [83.16 to 100.00]
  23F (n=21, 45, 20) | 100.00 [83.89 to 100.00] | 97.78 [88.23 to 99.94] | 100.00 [83.16 to 100.00]
  1 (n=21, 45, 20) | 100.00 [83.89 to 100.00] | 100.00 [92.13 to 100.00] | 100.00 [83.16 to 100.00]
  3 (n=21, 44, 20) | 95.24 [76.18 to 99.88] | 68.18 [52.42 to 81.39] | 50.00 [27.20 to 72.80]
  5 (n=21, 45, 20) | 100.00 [83.89 to 100.00] | 100.00 [92.13 to 100.00] | 100.00 [83.16 to 100.00]
  6A (n=21, 45, 20) | 100.00 [83.89 to 100.00] | 100.00 [92.13 to 100.00] | 100.00 [83.16 to 100.00]
  7F (n=21, 45, 20) | 100.00 [83.89 to 100.00] | 100.00 [92.13 to 100.00] | 100.00 [83.16 to 100.00]
  19A (n=21, 45, 20) | 100.00 [83.89 to 100.00] | 100.00 [92.13 to 100.00] | 100.00 [83.16 to 100.00]

20. Secondary Outcome: Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody Before Toddler Dose
Description: Geometric mean concentration (GMC) for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) were presented. GMC (13vPnC) and corresponding 2-sided 95% CI were evaluated. GMCs were calculated using all participants with available data for the specified blood draw. CIs were calculated as back transformations of a CI based on the Student t distribution for the mean logarithm of the concentrations.
Time Frame: Before Toddler Dose (pre-vaccination)
Population: Evaluable Toddler Immunogenicity Population. Here 'n' signifies participants with a determinate IgG concentration to the given serotype for each arm, respectively.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Number analyzed (Participants) | 88 | 88
mcg/mL
  4 (n= 85, 85) | 0.31 [0.26 to 0.37] | 0.41 [0.34 to 0.49]
  6B (n= 82, 85) | 0.48 [0.39 to 0.58] | 0.94 [0.79 to 1.11]
  9V (n= 85, 85) | 0.39 [0.33 to 0.46] | 0.62 [0.53 to 0.72]
  14 (n= 85, 85) | 2.02 [1.68 to 2.43] | 2.36 [1.94 to 2.87]
  18C (n=85, 85) | 0.32 [0.28 to 0.37] | 0.30 [0.26 to 0.36]
  19F (n=85, 85) | 0.68 [0.57 to 0.80] | 0.93 [0.79 to 1.10]
  23F (n=81, 83) | 0.24 [0.18 to 0.31] | 0.40 [0.33 to 0.48]
  1 (n=85, 85) | 0.39 [0.34 to 0.46] | 0.41 [0.35 to 0.48]
  3 (n=84, 84) | 0.07 [0.05 to 0.09] | 0.11 [0.09 to 0.14]
  5 (n=82, 85) | 0.74 [0.64 to 0.87] | 1.06 [0.90 to 1.26]
  6A (n=85, 85) | 0.54 [0.45 to 0.65] | 1.01 [0.82 to 1.24]
  7F (n=85, 85) | 0.72 [0.63 to 0.82] | 0.84 [0.73 to 0.96]
  19A (n=85, 85) | 0.86 [0.72 to 1.03] | 1.57 [1.27 to 1.92]
Statistical Analysis 1: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 4: Ratios of GMCs were calculated by back transforming the mean difference between vaccine groups on the logarithmic scale. CIs for the ratio were back transformations of a CI based on the Student t distribution for the ratio difference of the logarithms of the measures; Test type: Superiority or Other; GMC Ratio = 0.76, 95% CI 2-sided [0.60 to 0.97]
Statistical Analysis 2: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; GMC Ratio = 0.51, 95% CI 2-sided [0.39 to 0.66]
Statistical Analysis 3: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; GMC Ratio = 0.64, 95% CI 2-sided [0.51 to 0.80]
Statistical Analysis 4: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 14: Ratios of GMCs were calculated by back transforming the mean difference between vaccine groups on the logarithmic scale. CIs for the ratio were back transformations of a CI based on the Student t distribution for the ratio difference of the logarithms of the measures; Test type: Superiority or Other; GMC Ratio = 0.86, 95% CI 2-sided [0.66 to 1.12]
Statistical Analysis 5: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 18C: Ratios of GMCs were calculated by back transforming the mean difference between vaccine groups on the logarithmic scale. CIs for the ratio were back transformations of a CI based on the Student t distribution for the ratio difference of the logarithms of the measures; Test type: Superiority or Other; GMC Ratio = 1.06, 95% CI 2-sided [0.85 to 1.32]
Statistical Analysis 6: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 19F: Ratios of GMCs were calculated by back transforming the mean difference between vaccine groups on the logarithmic scale. CIs for the ratio were back transformations of a CI based on the Student t distribution for the ratio difference of the logarithms of the measures; Test type: Superiority or Other; GMC Ratio = 0.73, 95% CI 2-sided [0.58 to 0.92]
Statistical Analysis 7: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; GMC Ratio = 0.60, 95% CI 2-sided [0.43 to 0.83]
Statistical Analysis 8: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 8]; Test type: Superiority or Other; GMC Ratio = 0.96, 95% CI 2-sided [0.77 to 1.20]
Statistical Analysis 9: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; GMC Ratio = 0.60, 95% CI 2-sided [0.41 to 0.87]
Statistical Analysis 10: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 10]; Test type: Superiority or Other; GMC Ratio = 0.70, 95% CI 2-sided [0.56 to 0.88]
Statistical Analysis 11: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; GMC Ratio = 0.54, 95% CI 2-sided [0.41 to 0.70]
Statistical Analysis 12: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 12]; Test type: Superiority or Other; GMC Ratio = 0.86, 95% CI 2-sided [0.71 to 1.03]
Statistical Analysis 13: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 19A: Ratios of GMCs were calculated by back transforming the mean difference between vaccine groups on the logarithmic scale. CIs for the ratio were back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures; Test type: Superiority or Other; GMC Ratio = 0.55, 95% CI 2-sided [0.42 to 0.72]

21. Secondary Outcome: Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody 1 Month After Toddler Dose
Description: Geometric mean concentration (GMC) for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) were presented. GMC (13vPnC) and corresponding 2-sided 95% CI were evaluated. GMCs were calculated using all participants with available data for the specified blood draw. CIs were calculated as back transformations of a CI based on the Student t distribution for the mean logarithm of the concentrations. Here 'n' signifies participants with a determinate IgG concentration to the given serotype for each arm, respectively.
Time Frame: 1 Month After Toddler Dose
Population: Evaluable Toddler Immunogenicity Population.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Number analyzed (Participants) | 88 | 88
mcg/mL
  4 (n= 86, 87) | 2.57 [2.18 to 3.03] | 3.97 [3.32 to 4.74]
  6B (n=86, 87) | 4.42 [3.64 to 5.37] | 7.27 [6.09 to 8.68]
  9V (n=86, 87) | 2.30 [1.99 to 2.66] | 3.06 [2.62 to 3.56]
  14 (n=86, 87) | 9.24 [7.66 to 11.14] | 11.02 [9.44 to 12.86]
  18C (n=86, 87) | 2.37 [2.02 to 2.79] | 2.81 [2.32 to 3.40]
  19F (n=86, 87) | 7.38 [6.23 to 8.76] | 11.67 [9.47 to 14.36]
  23F (n=86, 87) | 2.45 [2.01 to 2.98] | 4.03 [3.36 to 4.85]
  1 (n=86, 87) | 3.32 [2.83 to 3.89] | 4.09 [3.42 to 4.89]
  3 (n=85, 87) | 0.52 [0.44 to 0.62] | 0.57 [0.49 to 0.65]
  5 (n=86, 87) | 2.63 [2.28 to 3.02] | 3.72 [3.19 to 4.33]
  6A (n=86, 87) | 5.64 [4.86 to 6.54] | 7.84 [6.59 to 9.33]
  7F (n=86, 87) | 4.25 [3.75 to 4.82] | 5.13 [4.48 to 5.87]
  19A (n=86, 87) | 5.57 [4.66 to 6.65] | 8.84 [7.45 to 10.48]
Statistical Analysis 1: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; GMC Ratio = 0.65, 95% CI 2-sided [0.51 to 0.82]
Statistical Analysis 2: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; GMC Ratio = 0.61, 95% CI 2-sided [0.47 to 0.79]
Statistical Analysis 3: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; GMC Ratio = 0.75, 95% CI 2-sided [0.61 to 0.93]
Statistical Analysis 4: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; GMC Ratio = 0.84, 95% CI 2-sided [0.66 to 1.07]
Statistical Analysis 5: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; GMC Ratio = 0.84, 95% CI 2-sided [0.66 to 1.08]
Statistical Analysis 6: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; GMC Ratio = 0.63, 95% CI 2-sided [0.48 to 0.83]
Statistical Analysis 7: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; GMC Ratio = 0.61, 95% CI 2-sided [0.46 to 0.79]
Statistical Analysis 8: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 8]; Test type: Superiority or Other; GMC Ratio = 0.81, 95% CI 2-sided [0.64 to 1.03]
Statistical Analysis 9: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; GMC Ratio = 0.92, 95% CI 2-sided [0.73 to 1.15]
Statistical Analysis 10: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 10]; Test type: Superiority or Other; GMC Ratio = 0.71, 95% CI 2-sided [0.58 to 0.87]
Statistical Analysis 11: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; GMC Ratio = 0.72, 95% CI 2-sided [0.57 to 0.90]
Statistical Analysis 12: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 12]; Test type: Superiority or Other; GMC Ratio = 0.83, 95% CI 2-sided [0.69 to 1.00]
Statistical Analysis 13: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 20, analysis 13]; Test type: Superiority or Other; GMC Ratio = 0.63, 95% CI 2-sided [0.49 to 0.81]

22. Secondary Outcome: Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody Persistence 1 Year After Toddler Dose
Description: The persistence of the antibody response induced by 13vPnC was described by geometric mean concentration (GMC) for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A). GMC (13vPnC) and corresponding 2-sided 95% CIs were evaluated. GMCs were calculated using all participants with available data for the specified blood draw. CIs were calculated as back transformations of a CI based on the Student t distribution for the mean logarithm of the concentrations.
Time Frame: 1 Year After Toddler Dose
Population: Evaluable Toddler Immunogenicity Population. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure during specified follow-up period and 'n' signifies participants with a determinate IgG concentration to the given serotype during specified follow-up period for each arm, respectively.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Number analyzed (Participants) | 80 | 80
mcg/mL
  4 (n= 80, 79) | 0.30 [0.25 to 0.36] | 0.37 [0.31 to 0.44]
  6B (n=80, 80) | 1.26 [1.02 to 1.57] | 2.01 [1.69 to 2.39]
  9V (n=80, 80) | 0.61 [0.48 to 0.78] | 0.98 [0.82 to 1.19]
  14 (n=79, 80) | 1.43 [1.15 to 1.78] | 1.73 [1.40 to 2.14]
  18C (n=80, 79) | 0.33 [0.27 to 0.41] | 0.66 [0.54 to 0.81]
  19F (n=80, 79) | 0.96 [0.80 to 1.15] | 1.78 [1.40 to 2.26]
  23F (n=79, 80) | 0.59 [0.47 to 0.74] | 1.24 [1.01 to 1.52]
  1 (n=78, 80) | 0.40 [0.35 to 0.46] | 0.53 [0.45 to 0.62]
  3 (n=78, 78) | 0.13 [0.10 to 0.17] | 0.22 [0.16 to 0.30]
  5 (n=79, 78) | 1.10 [0.91 to 1.32] | 1.63 [1.35 to 1.97]
  6A (n=80, 79) | 1.08 [0.89 to 1.32] | 1.59 [1.34 to 1.90]
  7F (n=79, 80) | 0.68 [0.59 to 0.80] | 0.83 [0.72 to 0.96]
  19A (n=80, 80) | 1.61 [1.22 to 2.12] | 3.16 [2.53 to 3.95]
Statistical Analysis 1: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; GMC Ratio = 0.81, 95% CI 2-sided [0.63 to 1.04]
Statistical Analysis 2: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; GMC Ratio = 0.63, 95% CI 2-sided [0.48 to 0.83]
Statistical Analysis 3: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; GMC Ratio = 0.62, 95% CI 2-sided [0.46 to 0.84]
Statistical Analysis 4: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; GMC Ratio = 0.83, 95% CI 2-sided [0.61 to 1.12]
Statistical Analysis 5: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; GMC Ratio = 0.50, 95% CI 2-sided [0.37 to 0.67]
Statistical Analysis 6: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; GMC Ratio = 0.54, 95% CI 2-sided [0.40 to 0.72]
Statistical Analysis 7: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; GMC Ratio = 0.47, 95% CI 2-sided [0.35 to 0.64]
Statistical Analysis 8: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 8]; Test type: Superiority or Other; GMC Ratio = 0.76, 95% CI 2-sided [0.61 to 0.94]
Statistical Analysis 9: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; GMC Ratio = 0.59, 95% CI 2-sided [0.39 to 0.90]
Statistical Analysis 10: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 10]; Test type: Superiority or Other; GMC Ratio = 0.67, 95% CI 2-sided [0.52 to 0.87]
Statistical Analysis 11: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; GMC Ratio = 0.68, 95% CI 2-sided [0.52 to 0.88]
Statistical Analysis 12: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 12]; Test type: Superiority or Other; GMC Ratio = 0.82, 95% CI 2-sided [0.67 to 1.02]
Statistical Analysis 13: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 20, analysis 13]; Test type: Superiority or Other; GMC Ratio = 0.51, 95% CI 2-sided [0.36 to 0.72]

23. Secondary Outcome: Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody Persistence 2 Years After Toddler Dose
Description: as for outcome 22
Time Frame: 2 Years After Toddler Dose
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Number analyzed (Participants) | 71 | 71
mcg/mL
  4 (n=70, 71) | 0.19 [0.16 to 0.23] | 0.24 [0.20 to 0.29]
  6B (n=70, 70) | 1.44 [1.13 to 1.85] | 2.70 [2.10 to 3.48]
  9V (n=71, 70) | 0.74 [0.58 to 0.94] | 0.99 [0.80 to 1.23]
  14 (n=70, 71) | 1.06 [0.78 to 1.43] | 1.37 [1.03 to 1.82]
  18C (n=69, 71) | 0.32 [0.24 to 0.42] | 0.57 [0.47 to 0.69]
  19F (n=71, 70) | 1.10 [0.83 to 1.46] | 2.43 [1.71 to 3.44]
  23F (n=71, 71) | 1.03 [0.77 to 1.38] | 1.83 [1.42 to 2.37]
  1 (n=70, 69) | 0.32 [0.26 to 0.38] | 0.39 [0.32 to 0.47]
  3 (n=65, 63) | 0.17 [0.12 to 0.25] | 0.27 [0.18 to 0.40]
  5 (n=69, 69) | 1.34 [1.07 to 1.68] | 1.97 [1.60 to 2.41]
  6A (n=71, 71) | 1.41 [1.09 to 1.82] | 2.10 [1.64 to 2.70]
  7F (n=71, 70) | 0.60 [0.50 to 0.71] | 0.67 [0.57 to 0.80]
  19A (n=71, 71) | 2.33 [1.76 to 3.10] | 4.36 [3.40 to 5.61]
Statistical Analysis 1: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; GMC Ratio = 0.80, 95% CI 2-sided [0.61 to 1.03]
Statistical Analysis 2: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; GMC Ratio = 0.53, 95% CI 2-sided [0.38 to 0.76]
Statistical Analysis 3: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; GMC Ratio = 0.74, 95% CI 2-sided [0.54 to 1.03]
Statistical Analysis 4: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; GMC Ratio = 0.77, 95% CI 2-sided [0.51 to 1.17]
Statistical Analysis 5: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; GMC Ratio = 0.56, 95% CI 2-sided [0.40 to 0.78]
Statistical Analysis 6: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; GMC Ratio = 0.45, 95% CI 2-sided [0.29 to 0.71]
Statistical Analysis 7: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; GMC Ratio = 0.56, 95% CI 2-sided [0.38 to 0.83]
Statistical Analysis 8: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 8]; Test type: Superiority or Other; GMC Ratio = 0.82, 95% CI 2-sided [0.63 to 1.07]
Statistical Analysis 9: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; GMC Ratio = 0.66, 95% CI 2-sided [0.39 to 1.11]
Statistical Analysis 10: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 10]; Test type: Superiority or Other; GMC Ratio = 0.68, 95% CI 2-sided [0.50 to 0.92]
Statistical Analysis 11: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; GMC Ratio = 0.67, 95% CI 2-sided [0.47 to 0.95]
Statistical Analysis 12: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 2, analysis 12]; Test type: Superiority or Other; GMC Ratio = 0.89, 95% CI 2-sided [0.70 to 1.13]
Statistical Analysis 13: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 20, analysis 13]; Test type: Superiority or Other; GMC Ratio = 0.53, 95% CI 2-sided [0.37 to 0.78]

24. Secondary Outcome: Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody 1 Month After Infant Series: Group 1A, 1B, 1C
Description: as for outcome 21
Time Frame: 1 Month After Infant Series
Population: Evaluable Infant Immunogenicity Population.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Groups:
- 13vPnC (Group 1C): Preterm participants with GA <29 weeks received single 0.5 mL dose of 13vPnC intramuscularly at 2, 3, 4 months of age (infant series) and at 12 months of age (toddler dose).
Arm/Group | 13vPnC (Group 1A) | 13vPnC (Group 1B) | 13vPnC (Group 1C)
Number analyzed (Participants) | 24 | 50 | 25
mcg/mL
  4 (n=24, 50, 25) | 2.50 [1.92 to 3.24] | 1.86 [1.47 to 2.37] | 1.73 [1.20 to 2.49]
  6B (n=24, 50, 25) | 1.23 [0.74 to 2.07] | 0.61 [0.42 to 0.88] | 0.62 [0.30 to 1.31]
  9V (n=24, 50, 25) | 1.44 [1.02 to 2.03] | 1.25 [1.02 to 1.53] | 1.14 [0.78 to 1.65]
  14 (n=24, 50, 25) | 8.95 [6.44 to 12.42] | 7.13 [5.65 to 8.98] | 6.95 [4.20 to 11.50]
  18C (n=24, 50, 25) | 2.58 [1.97 to 3.37] | 1.78 [1.44 to 2.19] | 1.72 [1.22 to 2.43]
  19F (n=24, 50, 25) | 2.46 [1.77 to 3.43] | 2.06 [1.67 to 2.55] | 2.28 [1.61 to 3.24]
  23F (n=24, 50, 25) | 1.38 [0.84 to 2.27] | 0.65 [0.48 to 0.89] | 0.95 [0.66 to 1.35]
  1 (n=24, 50, 25) | 1.56 [1.12 to 2.18] | 1.21 [0.96 to 1.52] | 1.10 [0.75 to 1.60]
  3 (n=24, 50, 25) | 1.28 [0.86 to 1.90] | 0.75 [0.60 to 0.93] | 0.67 [0.49 to 0.91]
  5 (n=24, 50, 25) | 0.85 [0.57 to 1.28] | 0.50 [0.36 to 0.69] | 0.46 [0.26 to 0.82]
  6A (n=24, 49, 25) | 1.74 [1.19 to 2.55] | 1.15 [0.84 to 1.57] | 0.98 [0.59 to 1.65]
  7F (n=24, 50, 25) | 2.43 [1.56 to 3.77] | 1.99 [1.61 to 2.46] | 2.18 [1.55 to 3.06]
  19A (n=24, 50, 25) | 3.43 [2.52 to 4.67] | 2.60 [2.08 to 3.25] | 2.88 [2.06 to 4.02]

25. Secondary Outcome: Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody Before Toddler Dose: Group 1A, 1B, 1C
Description: as for outcome 21
Time Frame: Before Toddler Dose (pre-vaccination)
Population: Evaluable Toddler Immunogenicity Population.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC (Group 1A) | 13vPnC (Group 1B) | 13vPnC (Group 1C)
Number analyzed (Participants) | 21 | 46 | 21
mcg/mL
  4 (n= 20, 44, 21) | 0.37 [0.27 to 0.50] | 0.28 [0.22 to 0.36] | 0.32 [0.22 to 0.46]
  6B (n= 20, 42, 20) | 0.59 [0.42 to 0.83] | 0.42 [0.31 to 0.56] | 0.49 [0.30 to 0.80]
  9V (n= 20, 44, 21) | 0.43 [0.30 to 0.60] | 0.36 [0.28 to 0.46] | 0.44 [0.33 to 0.60]
  14 (n=20, 44, 21) | 2.48 [1.74 to 3.54] | 1.83 [1.40 to 2.38] | 2.04 [1.33 to 3.12]
  18C (n=20, 44, 21) | 0.35 [0.25 to 0.48] | 0.30 [0.24 to 0.36] | 0.34 [0.24 to 0.49]
  19F (n=20, 44, 21) | 0.96 [0.57 to 1.61] | 0.58 [0.48 to 0.71] | 0.67 [0.52 to 0.87]
  23F (n=20, 41, 20) | 0.31 [0.19 to 0.52] | 0.21 [0.14 to 0.32] | 0.24 [0.14 to 0.41]
  1 (n=20, 44, 21) | 0.37 [0.27 to 0.52] | 0.39 [0.32 to 0.48] | 0.42 [0.30 to 0.61]
  3 (n=20, 44, 20) | 0.13 [0.07 to 0.24] | 0.06 [0.04 to 0.08] | 0.05 [0.02 to 0.09]
  5 (n=19, 43, 20) | 0.75 [0.56 to 1.01] | 0.71 [0.55 to 0.90] | 0.81 [0.62 to 1.06]
  6A (n=20, 44, 21) | 0.66 [0.46 to 0.93] | 0.49 [0.38 to 0.63] | 0.55 [0.35 to 0.85]
  7F (n=20, 44, 21) | 0.71 [0.55 to 0.92] | 0.64 [0.54 to 0.77] | 0.91 [0.69 to 1.19]
  19A (n=20, 44, 21) | 1.20 [0.76 to 1.89] | 0.72 [0.57 to 0.91] | 0.92 [0.66 to 1.30]

26. Secondary Outcome: Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody 1 Month After Toddler Dose: Group 1A, 1B, 1C
Description: as for outcome 21
Time Frame: 1 Month After Toddler Dose
Population: Evaluable Toddler Immunogenicity Population.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC (Group 1A) | 13vPnC (Group 1B) | 13vPnC (Group 1C)
Number analyzed (Participants) | 21 | 46 | 21
mcg/mL
  4 (n= 21, 45, 20) | 3.58 [2.66 to 4.83] | 2.87 [2.29 to 3.59] | 1.41 [1.05 to 1.88]
  6B (n= 21, 45, 20) | 6.28 [4.60 to 8.58] | 4.28 [3.18 to 5.75] | 3.29 [2.24 to 4.84]
  9V (n= 21, 45, 20) | 2.99 [2.26 to 3.96] | 2.23 [1.81 to 2.74] | 1.88 [1.41 to 2.52]
  14 (n=21, 45, 20) | 13.20 [9.65 to 18.05] | 8.84 [6.58 to 11.90] | 7.01 [5.15 to 9.54]
  18C (n=21, 45, 20) | 3.71 [2.77 to 4.97] | 2.40 [1.95 to 2.96] | 1.45 [1.05 to 2.00]
  19F (n=21, 45, 20) | 10.45 [8.20 to 13.32] | 7.39 [5.62 to 9.71] | 5.12 [3.91 to 6.72]
  23F (n=21, 45, 20) | 3.57 [2.54 to 5.02] | 2.41 [1.80 to 3.21] | 1.71 [1.12 to 2.62]
  1 (n=21, 45, 20) | 4.78 [3.61 to 6.34] | 3.31 [2.62 to 4.18] | 2.28 [1.74 to 2.99]
  3 (n=21, 44, 20) | 0.88 [0.61 to 1.25] | 0.51 [0.41 to 0.64] | 0.31 [0.23 to 0.43]
  5 (n=21, 45, 20) | 3.41 [2.69 to 4.32] | 2.66 [2.14 to 3.30] | 1.95 [1.54 to 2.47]
  6A (n=21, 45, 20) | 6.95 [5.18 to 9.33] | 5.81 [4.68 to 7.22] | 4.23 [3.22 to 5.56]
  7F (n=21, 45, 20) | 5.29 [4.11 to 6.80] | 4.09 [3.41 to 4.89] | 3.69 [2.84 to 4.80]
  19A (n=21, 45, 20) | 8.63 [6.51 to 11.43] | 5.28 [3.96 to 7.04] | 3.96 [3.17 to 4.96]

27. Secondary Outcome: Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody Persistence 1 Year After Toddler Dose: Group 1A, 1B, 1C
Description: as for outcome 22
Time Frame: 1 Year After Toddler Dose
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC (Group 1A) | 13vPnC (Group 1B) | 13vPnC (Group 1C)
Number analyzed (Participants) | 18 | 43 | 19
mcg/mL
  4 (n=18, 43, 19) | 0.30 [0.19 to 0.46] | 0.29 [0.23 to 0.37] | 0.32 [0.21 to 0.49]
  6B (n=18, 43, 19) | 1.49 [0.84 to 2.66] | 1.28 [0.96 to 1.70] | 1.06 [0.70 to 1.60]
  9V (n=18, 43, 19) | 0.59 [0.37 to 0.93] | 0.56 [0.42 to 0.75] | 0.80 [0.40 to 1.59]
  14 (n=18, 42, 19) | 1.37 [0.86 to 2.19] | 1.38 [1.09 to 1.75] | 1.62 [0.83 to 3.16]
  18C (n=18, 43, 19) | 0.39 [0.26 to 0.57] | 0.31 [0.24 to 0.41] | 0.32 [0.17 to 0.59]
  19F (n=18, 43, 19) | 1.27 [0.81 to 2.00] | 0.89 [0.70 to 1.14] | 0.86 [0.62 to 1.21]
  23F (n=18, 42, 19) | 0.79 [0.50 to 1.26] | 0.54 [0.40 to 0.74] | 0.53 [0.30 to 0.91]
  1 (n=18, 41, 19) | 0.39 [0.30 to 0.50] | 0.38 [0.32 to 0.47] | 0.45 [0.31 to 0.64]
  3 (n=18, 41, 19) | 0.17 [0.10 to 0.29] | 0.12 [0.09 to 0.17] | 0.11 [0.05 to 0.23]
  5 (n=18, 42, 19) | 0.87 [0.59 to 1.28] | 1.24 [0.93 to 1.64] | 1.05 [0.77 to 1.44]
  6A (n=18, 43, 19) | 1.17 [0.73 to 1.87] | 1.05 [0.80 to 1.40] | 1.07 [0.72 to 1.59]
  7F (n=18, 42, 19) | 0.65 [0.47 to 0.91] | 0.65 [0.52 to 0.81] | 0.81 [0.61 to 1.08]
  19A (n=18, 43, 19) | 2.12 [0.90 to 5.01] | 1.50 [1.05 to 2.14] | 1.45 [0.95 to 2.21]

28. Secondary Outcome: Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody Persistence 2 Years After Toddler Dose: Group 1A, 1B, 1C
Description: as for outcome 22
Time Frame: 2 Years After Toddler Dose
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC (Group 1A) | 13vPnC (Group 1B) | 13vPnC (Group 1C)
Number analyzed (Participants) | 17 | 36 | 18
mcg/mL
  4 (n=17, 35, 18) | 0.17 [0.11 to 0.28] | 0.19 [0.16 to 0.24] | 0.21 [0.13 to 0.33]
  6B (n=17, 35, 18) | 1.39 [0.81 to 2.40] | 1.81 [1.28 to 2.56] | 0.96 [0.58 to 1.60]
  9V (n=17, 36, 18) | 0.68 [0.39 to 1.17] | 0.83 [0.59 to 1.16] | 0.63 [0.36 to 1.12]
  14 (n=17, 35, 18) | 1.27 [0.59 to 2.76] | 1.02 [0.71 to 1.48] | 0.96 [0.47 to 1.96]
  18C (n=16, 35, 18) | 0.34 [0.18 to 0.65] | 0.35 [0.23 to 0.52] | 0.26 [0.16 to 0.44]
  19F (n=17, 36, 18) | 1.53 [0.83 to 2.81] | 0.93 [0.68 to 1.28] | 1.13 [0.50 to 2.53]
  23F (n=17, 36, 18) | 1.14 [0.60 to 2.15] | 1.41 [0.95 to 2.09] | 0.50 [0.27 to 0.90]
  1 (n=17, 35, 18) | 0.32 [0.23 to 0.44] | 0.35 [0.26 to 0.47] | 0.26 [0.18 to 0.39]
  3 (n=16, 33, 16) | 0.20 [0.10 to 0.39] | 0.19 [0.11 to 0.30] | 0.14 [0.06 to 0.34]
  5 (n=17, 35, 17) | 1.18 [0.67 to 2.11] | 1.67 [1.25 to 2.25] | 0.97 [0.62 to 1.50]
  6A (n=17, 36, 18) | 1.32 [0.87 to 1.99] | 1.58 [1.10 to 2.26] | 1.20 [0.63 to 2.30]
  7F (n=17, 36, 18) | 0.61 [0.39 to 0.96] | 0.68 [0.54 to 0.84] | 0.46 [0.32 to 0.67]
  19A (n=17, 36, 18) | 3.04 [1.64 to 5.64] | 2.46 [1.69 to 3.58] | 1.64 [0.83 to 3.23]

29. Secondary Outcome: Serotype-Specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titer (GMT) 1 Month After Infant Series
Description: Antibody-mediated serum OPA against the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) was measured centrally using a pneumococcal OPA assay. Results were expressed as OPA titers. OPA titers were logarithmically transformed for analysis; geometric means calculated and expressed as geometric mean titers (GMTs).
Time Frame: 1 Month After Infant Series
Population: Evaluable Infant Immunogenicity Population. Here n' signifies participants with a determinate OPA titer to the given serotype for each arm respectively.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Number analyzed (Participants) | 99 | 98
titer
  4 (n=58, 62) | 1231 [986.5 to 1537.3] | 923 [746.9 to 1139.7]
  6B (n=51, 61) | 835 [478.6 to 1455.2] | 732 [494.0 to 1086.0]
  9V (n=54, 60) | 151 [70.8 to 321.1] | 211 [108.2 to 413.4]
  14 (n=55, 66) | 1298 [968.3 to 1740.3] | 1033 [735.7 to 1451.0]
  18C (n=56, 63) | 2931 [2341.2 to 3669.3] | 2057 [1594.0 to 2655.1]
  19F (n= 55, 58) | 417 [330.7 to 525.8] | 335 [237.2 to 472.3]
  23F (n=55, 60) | 733 [539.3 to 997.3] | 582 [413.7 to 817.8]
  1 (n=88, 87) | 10 [8.0 to 13.4] | 13 [10.0 to 16.8]
  3 (n=83, 86) | 61 [51.2 to 73.2] | 57 [46.3 to 69.5]
  5 (n=83, 85) | 37 [25.9 to 53.9] | 64 [47.2 to 86.9]
  6A (n=88, 88) | 1566 [1312.3 to 1869.0] | 1287 [980.1 to 1691.1]
  7F (n=93, 86) | 1605 [1277.9 to 2014.7] | 1539 [1297.4 to 1826.3]
  19A (n=92, 86) | 283 [232.4 to 344.1] | 244 [204.1 to 290.6]
Statistical Analysis 1: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 4: Ratio of GMTs calculated by back transforming the mean difference between the groups on the logarithmic scale. CIs for the ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures; Test type: Superiority or Other; GMT Ratio = 1.3, 95% CI 2-sided [0.99 to 1.81]
Statistical Analysis 2: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 6B: Ratio of GMTs calculated by back transforming the mean difference between the groups on the logarithmic scale. CIs for the ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures; Test type: Superiority or Other; GMT Ratio = 1.1, 95% CI 2-sided [0.59 to 2.20]
Statistical Analysis 3: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 9V: Ratio of GMTs calculated by back transforming the mean difference between the groups on the logarithmic scale. CIs for the ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures; Test type: Superiority or Other; GMT Ratio = 0.7, 95% CI 2-sided [0.26 to 1.93]
Statistical Analysis 4: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 14: Ratio of GMTs calculated by back transforming the mean difference between the groups on the logarithmic scale. CIs for the ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures; Test type: Superiority or Other; GMT Ratio = 1.3, 95% CI 2-sided [0.80 to 1.98]
Statistical Analysis 5: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 18C: Ratio of GMTs calculated by back transforming the mean difference between the groups on the logarithmic scale. CIs for the ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures; Test type: Superiority or Other; GMT Ratio = 1.4, 95% CI 2-sided [1.01 to 2.00]
Statistical Analysis 6: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 19F: Ratio of GMTs calculated by back transforming the mean difference between the groups on the logarithmic scale. CIs for the ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures; Test type: Superiority or Other; GMT Ratio = 1.2, 95% CI 2-sided [0.82 to 1.89]
Statistical Analysis 7: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 23F: Ratio of GMTs calculated by back transforming the mean difference between the groups on the logarithmic scale. CIs for the ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures; Test type: Superiority or Other; GMT Ratio = 1.3, 95% CI 2-sided [0.80 to 1.99]
Statistical Analysis 8: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 1: Ratio of GMTs calculated by back transforming the mean difference between the groups on the logarithmic scale. CIs for the ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures; Test type: Superiority or Other; GMT Ratio = 0.8, 95% CI 2-sided [0.56 to 1.15]
Statistical Analysis 9: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 3: Ratio of GMTs calculated by back transforming the mean difference between the groups on the logarithmic scale. CIs for the ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures; Test type: Superiority or Other; GMT Ratio = 1.1, 95% CI 2-sided [0.83 to 1.41]
Statistical Analysis 10: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 5: Ratio of GMTs calculated by back transforming the mean difference between the groups on the logarithmic scale. CIs for the ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures; Test type: Superiority or Other; GMT Ratio = 0.6, 95% CI 2-sided [0.36 to 0.94]
Statistical Analysis 11: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 6A: Ratio of GMTs calculated by back transforming the mean difference between the groups on the logarithmic scale. CIs for the ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures; Test type: Superiority or Other; GMT Ratio = 1.2, 95% CI 2-sided [0.88 to 1.68]
Statistical Analysis 12: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 7F: Ratio of GMTs calculated by back transforming the mean difference between the groups on the logarithmic scale. CIs for the ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures; Test type: Superiority or Other; GMT Ratio = 1.0, 95% CI 2-sided [0.78 to 1.39]
Statistical Analysis 13: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 19A: Ratio of GMTs calculated by back transforming the mean difference between the groups on the logarithmic scale. CIs for the ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures; Test type: Superiority or Other; GMT Ratio = 1.2, 95% CI 2-sided [0.89 to 1.51]

30. Secondary Outcome: Serotype-Specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titer (GMT) Before Toddler Dose
Description: as for outcome 29
Time Frame: Before the toddler dose (pre-vaccination)
Population: Evaluable Toddler Immunogenicity Population. Here 'n' signifies participants with a determinate OPA titer to the given serotype for each arm respectively.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Number analyzed (Participants) | 88 | 88
titer
  4 (n= 56, 59) | 10 [6.0 to 15.3] | 13 [7.9 to 21.9]
  6B (n= 59, 62) | 12 [6.8 to 20.1] | 15 [8.5 to 25.6]
  9V (n=52, 63) | 11 [6.2 to 20.9] | 7 [4.9 to 11.1]
  14 (n= 60, 55) | 242 [148.5 to 394.0] | 389 [260.4 to 582.2]
  18C (n= 54, 58) | 32 [16.1 to 61.7] | 51 [26.8 to 98.3]
  19F (n= 57, 60) | 6 [4.1 to 7.4] | 4 [3.8 to 4.7]
  23F (n=59, 62) | 11 [6.9 to 19.0] | 16 [9.6 to 26.6]
  1 (n=76, 80) | 6 [4.5 to 6.8] | 4 [3.9 to 4.8]
  3 (n=73, 77) | 8 [6.2 to 10.0] | 8 [6.6 to 10.4]
  5 (n=74, 79) | 5 [4.2 to 6.0] | 5 [4.2 to 5.6]
  6A (n=69, 76) | 45 [25.2 to 81.1] | 91 [56.6 to 146.3]
  7F (n=75, 79) | 228 [137.6 to 377.1] | 188 [109.3 to 323.1]
  19A (n=77, 79) | 9 [6.3 to 12.0] | 10 [7.1 to 14.8]
Statistical Analysis 1: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 1]; Test type: Superiority or Other; GMT Ratio = 0.7, 95% CI 2-sided [0.37 to 1.44]
Statistical Analysis 2: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 2]; Test type: Superiority or Other; GMT Ratio = 0.8, 95% CI 2-sided [0.37 to 1.71]
Statistical Analysis 3: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 3]; Test type: Superiority or Other; GMT Ratio = 1.5, 95% CI 2-sided [0.76 to 3.12]
Statistical Analysis 4: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 4]; Test type: Superiority or Other; GMT Ratio = 0.6, 95% CI 2-sided [0.33 to 1.17]
Statistical Analysis 5: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 5]; Test type: Superiority or Other; GMT Ratio = 0.6, 95% CI 2-sided [0.24 to 1.55]
Statistical Analysis 6: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 6]; Test type: Superiority or Other; GMT Ratio = 1.3, 95% CI 2-sided [0.97 to 1.77]
Statistical Analysis 7: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 7]; Test type: Superiority or Other; GMT Ratio = 0.7, 95% CI 2-sided [0.35 to 1.46]
Statistical Analysis 8: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 8]; Test type: Superiority or Other; GMT Ratio = 1.3, 95% CI 2-sided [1.00 to 1.60]
Statistical Analysis 9: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 9]; Test type: Superiority or Other; GMT Ratio = 1.0, 95% CI 2-sided [0.68 to 1.33]
Statistical Analysis 10: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 10]; Test type: Superiority or Other; GMT Ratio = 1.0, 95% CI 2-sided [0.82 to 1.31]
Statistical Analysis 11: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 11]; Test type: Superiority or Other; GMT Ratio = 0.5, 95% CI 2-sided [0.24 to 1.04]
Statistical Analysis 12: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 12]; Test type: Superiority or Other; GMT Ratio = 1.2, 95% CI 2-sided [0.58 to 2.53]
Statistical Analysis 13: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 13]; Test type: Superiority or Other; GMT Ratio = 0.8, 95% CI 2-sided [0.52 to 1.37]

31. Secondary Outcome: Serotype-Specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titer (GMT) 1 Month After Toddler Dose
Description: as for outcome 29
Time Frame: 1 Month After Toddler Dose
Population: as for outcome 30
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Number analyzed (Participants) | 88 | 88
titer
  4 (n= 67, 61) | 1154 [879.2 to 1514.5] | 1757 [1329.1 to 2322.4]
  6B (n= 64, 61) | 1229 [877.2 to 1722.1] | 1406 [1003.4 to 1970.3]
  9V (n=60, 58) | 1871 [1217.8 to 2873.6] | 2542 [1711.6 to 3775.2]
  14 (n= 62, 62) | 1294 [969.0 to 1728.4] | 1651 [1300.1 to 2097.1]
  18C (n= 62, 63) | 2464 [1696.0 to 3579.4] | 4510 [3399.7 to 5981.7]
  19F (n= 61, 62) | 376 [229.1 to 617.1] | 640 [431.5 to 948.3]
  23F (n=65, 63) | 1048 [738.6 to 1488.0] | 1657 [1217.7 to 2255.0]
  1 (n=80, 83) | 59 [43.7 to 78.6] | 107 [83.0 to 137.0]
  3 (n=78, 79) | 114 [97.1 to 132.7] | 121 [103.4 to 140.4]
  5 (n=80, 83) | 166 [127.9 to 216.3] | 260 [203.9 to 331.9]
  6A (n=78, 74) | 1978 [1571.5 to 2489.7] | 3154 [2606.0 to 3816.0]
  7F (n=81, 82) | 2915 [2453.4 to 3462.7] | 3154 [2746.2 to 3622.4]
  19A (n=81, 82) | 558 [456.3 to 682.6] | 825 [692.4 to 983.8]
Statistical Analysis 1: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 1]; Test type: Superiority or Other; GMT Ratio = 0.7, 95% CI 2-sided [0.45 to 0.97]
Statistical Analysis 2: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 2]; Test type: Superiority or Other; GMT Ratio = 0.9, 95% CI 2-sided [0.54 to 1.40]
Statistical Analysis 3: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 3]; Test type: Superiority or Other; GMT Ratio = 0.7, 95% CI 2-sided [0.41 to 1.31]
Statistical Analysis 4: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 4]; Test type: Superiority or Other; GMT Ratio = 0.8, 95% CI 2-sided [0.54 to 1.14]
Statistical Analysis 5: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 5]; Test type: Superiority or Other; GMT Ratio = 0.5, 95% CI 2-sided [0.34 to 0.87]
Statistical Analysis 6: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 6]; Test type: Superiority or Other; GMT Ratio = 0.6, 95% CI 2-sided [0.31 to 1.10]
Statistical Analysis 7: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 7]; Test type: Superiority or Other; GMT Ratio = 0.6, 95% CI 2-sided [0.40 to 1.01]
Statistical Analysis 8: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 8]; Test type: Superiority or Other; GMT Ratio = 0.5, 95% CI 2-sided [0.38 to 0.81]
Statistical Analysis 9: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 9]; Test type: Superiority or Other; GMT Ratio = 0.9, 95% CI 2-sided [0.76 to 1.17]
Statistical Analysis 10: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 10]; Test type: Superiority or Other; GMT Ratio = 0.6, 95% CI 2-sided [0.45 to 0.91]
Statistical Analysis 11: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 11]; Test type: Superiority or Other; GMT Ratio = 0.6, 95% CI 2-sided [0.47 to 0.85]
Statistical Analysis 12: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 12]; Test type: Superiority or Other; GMT Ratio = 0.9, 95% CI 2-sided [0.74 to 1.15]
Statistical Analysis 13: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 13]; Test type: Superiority or Other; GMT Ratio = 0.7, 95% CI 2-sided [0.52 to 0.88]

32. Secondary Outcome: Serotype-Specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titer (GMT) 1 Year After Toddler Dose
Description: as for outcome 29
Time Frame: 1 Year After Toddler Dose
Population: Evaluable Toddler Immunogenicity Population. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure during specified follow-up period and 'n' signifies participants with a determinate OPA titer to the given serotype during specified follow-up period for each arm, respectively.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Number analyzed (Participants) | 80 | 80
titer
  4 (n= 66, 59) | 24 [12.9 to 45.5] | 29 [15.2 to 54.5]
  6B (n= 65, 59) | 38 [19.0 to 74.9] | 36 [19.2 to 68.8]
  9V (n=61, 63) | 141 [67.5 to 293.1] | 244 [126.3 to 469.7]
  14 (n= 59, 54) | 276 [169.0 to 449.4] | 372 [236.1 to 586.5]
  18C (n= 62, 60) | 33 [16.4 to 67.4] | 121 [56.9 to 258.1]
  19F (n= 67, 57) | 11 [6.2 to 17.7] | 18 [9.6 to 35.4]
  23F (n=67, 62) | 45 [23.7 to 86.6] | 168 [92.4 to 303.9]
  1 (n=76, 74) | 5 [4.2 to 6.3] | 5 [4.3 to 5.8]
  3 (n=76, 70) | 11 [8.6 to 15.4] | 13 [9.2 to 18.7]
  5 (n=72, 70) | 8 [5.6 to 10.4] | 10 [7.0 to 13.3]
  6A (n=70, 70) | 98 [53.0 to 183.0] | 255 [152.9 to 424.8]
  7F (n=71, 71) | 599 [411.0 to 873.3] | 533 [348.3 to 814.1]
  19A (n=74, 73) | 28 [17.2 to 43.9] | 54 [34.2 to 85.5]
Statistical Analysis 1: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 1]; Test type: Superiority or Other; GMT Ratio = 0.8, 95% CI 2-sided [0.35 to 2.05]
Statistical Analysis 2: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 2]; Test type: Superiority or Other; GMT Ratio = 1.0, 95% CI 2-sided [0.41 to 2.63]
Statistical Analysis 3: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 3]; Test type: Superiority or Other; GMT Ratio = 0.6, 95% CI 2-sided [0.22 to 1.53]
Statistical Analysis 4: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 4]; Test type: Superiority or Other; GMT Ratio = 0.7, 95% CI 2-sided [0.38 to 1.44]
Statistical Analysis 5: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 5]; Test type: Superiority or Other; GMT Ratio = 0.3, 95% CI 2-sided [0.10 to 0.76]
Statistical Analysis 6: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 6]; Test type: Superiority or Other; GMT Ratio = 0.6, 95% CI 2-sided [0.25 to 1.30]
Statistical Analysis 7: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 7]; Test type: Superiority or Other; GMT Ratio = 0.3, 95% CI 2-sided [0.11 to 0.65]
Statistical Analysis 8: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 8]; Test type: Superiority or Other; GMT Ratio = 1.0, 95% CI 2-sided [0.81 to 1.32]
Statistical Analysis 9: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 9]; Test type: Superiority or Other; GMT Ratio = 0.9, 95% CI 2-sided [0.56 to 1.37]
Statistical Analysis 10: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 10]; Test type: Superiority or Other; GMT Ratio = 0.8, 95% CI 2-sided [0.51 to 1.23]
Statistical Analysis 11: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 11]; Test type: Superiority or Other; GMT Ratio = 0.4, 95% CI 2-sided [0.17 to 0.86]
Statistical Analysis 12: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 12]; Test type: Superiority or Other; GMT Ratio = 1.1, 95% CI 2-sided [0.64 to 1.97]
Statistical Analysis 13: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 13]; Test type: Superiority or Other; GMT Ratio = 0.5, 95% CI 2-sided [0.27 to 0.97]

33. Secondary Outcome: Serotype-Specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titer (GMT) 2 Years After Toddler Dose
Description: Antibody-mediated serum OPA against the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) was measured using a pneumococcal OPA assay. Results were expressed as OPA titers. OPA titers were logarithmically transformed for analysis; geometric means calculated and expressed as geometric mean titers (GMTs).
Time Frame: 2 Years After Toddler Dose
Population: as for outcome 32
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Number analyzed (Participants) | 71 | 71
titer
  4 (n= 46, 54) | 15 [7.0 to 32.9] | 17 [9.0 to 32.6]
  6B (n= 56, 48) | 29 [13.7 to 59.9] | 27 [12.4 to 58.2]
  9V (n=50, 55) | 132 [57.5 to 301.5] | 75 [34.7 to 163.7]
  14 (n= 49, 45) | 262 [142.0 to 482.8] | 296 [161.6 to 543.8]
  18C (n= 56, 56) | 14 [7.1 to 25.9] | 29 [14.3 to 57.9]
  19F (n= 60, 58) | 13 [7.4 to 22.5] | 20 [10.1 to 39.9]
  23F (n=58, 59) | 60 [29.7 to 122.2] | 135 [71.2 to 255.3]
  1 (n=70, 68) | 5 [4.1 to 5.4] | 4 [3.9 to 4.6]
  3 (n=69, 66) | 11 [8.1 to 15.2] | 16 [10.7 to 24.2]
  5 (n=68, 69) | 5 [4.1 to 5.6] | 7 [5.4 to 9.4]
  6A (n=68, 62) | 42 [21.5 to 81.1] | 102 [53.7 to 193.4]
  7F (n=64, 65) | 170 [87.7 to 330.9] | 269 [155.6 to 463.7]
  19A (n=68, 67) | 22 [13.6 to 37.1] | 50 [30.1 to 82.6]
Statistical Analysis 1: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 1]; Test type: Superiority or Other; GMT Ratio = 0.9, 95% CI 2-sided [0.33 to 2.37]
Statistical Analysis 2: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 2]; Test type: Superiority or Other; GMT Ratio = 1.1, 95% CI 2-sided [0.37 to 3.07]
Statistical Analysis 3: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 3]; Test type: Superiority or Other; GMT Ratio = 1.7, 95% CI 2-sided [0.57 to 5.36]
Statistical Analysis 4: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 4]; Test type: Superiority or Other; GMT Ratio = 0.9, 95% CI 2-sided [0.38 to 2.07]
Statistical Analysis 5: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 5]; Test type: Superiority or Other; GMT Ratio = 0.5, 95% CI 2-sided [0.18 to 1.21]
Statistical Analysis 6: Comparison: 13vPnC Group 1 (Preterm Infant); [analysis description as in outcome 29, analysis 6]; Test type: Superiority or Other; GMT Ratio = 0.6, 95% CI 2-sided [0.27 to 1.53]
Statistical Analysis 7: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 7]; Test type: Superiority or Other; GMT Ratio = 0.4, 95% CI 2-sided [0.17 to 1.15]
Statistical Analysis 8: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 8]; Test type: Superiority or Other; GMT Ratio = 1.1, 95% CI 2-sided [0.96 to 1.31]
Statistical Analysis 9: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 9]; Test type: Superiority or Other; GMT Ratio = 0.7, 95% CI 2-sided [0.41 to 1.14]
Statistical Analysis 10: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 10]; Test type: Superiority or Other; GMT Ratio = 0.7, 95% CI 2-sided [0.49 to 0.92]
Statistical Analysis 11: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 11]; Test type: Superiority or Other; GMT Ratio = 0.4, 95% CI 2-sided [0.16 to 1.03]
Statistical Analysis 12: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 12]; Test type: Superiority or Other; GMT Ratio = 0.6, 95% CI 2-sided [0.27 to 1.48]
Statistical Analysis 13: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 29, analysis 13]; Test type: Superiority or Other; GMT Ratio = 0.5, 95% CI 2-sided [0.22 to 0.91]

34. Secondary Outcome: Percentage of Participants With OPA Titer >= Lower Limit of Quantitation (LLOQ) 1 Month After Infant Series
Description: Percentage of participants achieving OPA titer >=LLOQ for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) determined in blood samples of all participants was presented. Exact 2-sided CI based on observed proportion of participants. LLOQ for each serotype: 1=18; 3=12; 4=21; 5=29; 6A=37; 6B=43; 7F=210; 9V=345; 14=35; 18C=31; 19A=18; 19F=48; 23F=13.
Time Frame: 1 Month After Infant Series
Population: Evaluable Infant Immunogenicity Population. Here 'n' signifies participants with a determinate OPA antibody titer to the given serotype for each arm respectively.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Number analyzed (Participants) | 99 | 98
percentage of participants
  4 (n= 58, 62) | 100.00 [93.84 to 100.00] | 100.00 [94.22 to 100.00]
  6B (n= 51, 61) | 90.20 [78.59 to 96.74] | 95.08 [86.29 to 98.97]
  9V (n= 54, 60) | 64.81 [50.62 to 77.32] | 71.67 [58.56 to 82.55]
  14 (n= 55, 66) | 100.00 [93.51 to 100.00] | 96.97 [89.48 to 99.63]
  18C (n= 56, 63) | 100.00 [93.62 to 100.00] | 100.00 [94.31 to 100.00]
  19F (n= 55, 58) | 100.00 [93.51 to 100.00] | 96.55 [88.09 to 99.58]
  23F (n= 55, 60) | 98.18 [90.28 to 99.95] | 96.67 [88.47 to 99.59]
  1 (n= 88, 87) | 40.91 [30.54 to 51.91] | 51.72 [40.75 to 62.58]
  3 (n=83, 86) | 100.00 [95.65 to 100.00] | 95.35 [88.52 to 98.72]
  5 (n= 83, 85) | 67.47 [56.30 to 77.35] | 83.53 [73.91 to 90.69]
  6A (n= 88, 88) | 100.00 [95.89 to 100.00] | 97.73 [92.03 to 99.72]
  7F (n= 93, 86) | 97.85 [92.45 to 99.74] | 100.00 [95.80 to 100.00]
  19A (n= 92, 86) | 98.91 [94.09 to 99.97] | 100.00 [95.80 to 100.00]
Statistical Analysis 1: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 4: Exact 2-sided, 95% CI was computed based on the procedure of Chan and Zhang using the standardized test statistics and gamma=0.000001; Test type: Superiority or Other; Percent Difference = 0.00, 95% CI 2-sided [-6.33 to 5.99]
Statistical Analysis 2: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 6B: Exact 2-sided, 95% CI was computed based on the procedure of Chan and Zhang using the standardized test statistics and gamma=0.000001; Test type: Superiority or Other; Percent Difference = -4.89, 95% CI 2-sided [-16.87 to 5.39]
Statistical Analysis 3: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 9V: Exact 2-sided, 95% CI was computed based on the procedure of Chan and Zhang using the standardized test statistics and gamma=0.000001; Test type: Superiority or Other; Percent Difference = -6.85, 95% CI 2-sided [-24.28 to 10.67]
Statistical Analysis 4: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 14: Exact 2-sided, 95% CI was computed based on the procedure of Chan and Zhang using the standardized test statistics and gamma=0.000001; Test type: Superiority or Other; Percent Difference = 3.03, 95% CI 2-sided [-3.68 to 10.57]
Statistical Analysis 5: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 18C: Exact 2-sided, 95% CI was computed based on the procedure of Chan and Zhang using the standardized test statistics and gamma=0.000001; Test type: Superiority or Other; Percent Difference = 0.00, 95% CI 2-sided [-6.57 to 5.88]
Statistical Analysis 6: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 19F: Exact 2-sided, 95% CI was computed based on the procedure of Chan and Zhang using the standardized test statistics and gamma=0.000001; Test type: Superiority or Other; Percent Difference = 3.45, 95% CI 2-sided [-3.32 to 11.91]
Statistical Analysis 7: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 23F: Exact 2-sided, 95% CI was computed based on the procedure of Chan and Zhang using the standardized test statistics and gamma=0.000001; Test type: Superiority or Other; Percent Difference = 1.52, 95% CI 2-sided [-6.73 to 9.94]
Statistical Analysis 8: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 1: Exact 2-sided, 95% CI was computed based on the procedure of Chan and Zhang using the standardized test statistics and gamma=0.000001; Test type: Superiority or Other; Perecent Difference = -10.82, 95% CI 2-sided [-25.51 to 4.34]
Statistical Analysis 9: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 3: Exact 2-sided, 95% CI was computed based on the procedure of Chan and Zhang using the standardized test statistics and gamma=0.000001; Test type: Superiority or Other; Percent Difference = 4.65, 95% CI 2-sided [0.04 to 11.48]
Statistical Analysis 10: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 5: Exact 2-sided, 95% CI was computed based on the procedure of Chan and Zhang using the standardized test statistics and gamma=0.000001; Test type: Superiority or Other; Percent Difference = -16.06, 95% CI 2-sided [-29.15 to -2.60]
Statistical Analysis 11: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 6A: Exact 2-sided, 95% CI was computed based on the procedure of Chan and Zhang using the standardized test statistics and gamma=0.000001; Test type: Superiority or Other; Percent Difference = 2.27, 95% CI 2-sided [-1.96 to 7.97]
Statistical Analysis 12: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 7F: Exact 2-sided, 95% CI was computed based on the procedure of Chan and Zhang using the standardized test statistics and gamma=0.000001; Test type: Superiority or Other; Percent Difference = -2.15, 95% CI 2-sided [-7.55 to 2.10]
Statistical Analysis 13: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 19A: Exact 2-sided, 95% CI was computed based on the procedure of Chan and Zhang using the standardized test statistics and gamma=0.000001; Test type: Superiority or Other; Percent Difference = -1.09, 95% CI 2-sided [-5.96 to 3.18]

35. Secondary Outcome: Percentage of Participants With OPA Titer >= Lower Limit of Quantitation (LLOQ) Before Toddler Dose
Description: as for outcome 34
Time Frame: Before Toddler Dose (pre-vaccination)
Population: Evaluable Toddler Immunogenicity Population. Here 'n' signifies participants with a determinate OPA antibody titer to the given serotype for each arm respectively.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Number analyzed (Participants) | 88 | 88
percentage of participants
  4 (n=56, 59) | 21.43 [11.59 to 34.44] | 30.51 [19.19 to 43.87]
  6B (n=59, 62) | 22.03 [12.29 to 34.73] | 27.42 [16.85 to 40.23]
  9V (n=52, 63) | 19.23 [9.63 to 32.53] | 12.70 [5.65 to 23.50]
  14 (n=60, 55) | 86.67 [75.41 to 94.06] | 94.55 [84.88 to 98.86]
  18C (n=54, 58) | 44.44 [30.92 to 58.60] | 55.17 [41.54 to 68.26]
  19F (n=57, 60) | 8.77 [2.91 to 19.30] | 1.67 [0.04 to 8.94]
  23F (n=59, 62) | 23.73 [13.62 to 36.59] | 37.10 [25.16 to 50.31]
  1 (n=76, 80) | 11.84 [5.56 to 21.29] | 3.75 [0.78 to 10.57]
  3 (n=73, 77) | 32.88 [22.33 to 44.87] | 40.26 [29.23 to 52.06]
  5 (n=74, 79) | 8.11 [3.03 to 16.82] | 7.59 [2.84 to 15.80]
  6A (n=69, 76) | 52.17 [39.80 to 64.35] | 72.37 [60.91 to 82.01]
  7F (n=75, 79) | 78.67 [67.68 to 87.29] | 73.42 [62.28 to 82.73]
  19A (n=77, 79) | 25.97 [16.64 to 37.23] | 29.11 [19.43 to 40.42]
Statistical Analysis 1: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 1]; Test type: Superiority or Other; Percent Difference = -9.08, 95% CI 2-sided [-25.11 to 7.49]
Statistical Analysis 2: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 2]; Test type: Superiority or Other; Percent Difference = -5.39, 95% CI 2-sided [-21.03 to 10.40]
Statistical Analysis 3: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 3]; Test type: Superiority or Other; Percent Difference = 6.53, 95% CI 2-sided [-7.16 to 21.16]
Statistical Analysis 4: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 4]; Test type: Superiority or Other; Percent Difference = -7.88, 95% CI 2-sided [-20.28 to 3.35]
Statistical Analysis 5: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 5]; Test type: Superiority or Other; Percent Difference = -10.73, 95% CI 2-sided [-29.01 to 8.11]
Statistical Analysis 6: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 6]; Test type: Superiority or Other; Percent Difference = 7.11, 95% CI 2-sided [-1.52 to 17.65]
Statistical Analysis 7: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 7]; Test type: Superiority or Other; Percent Difference = -13.37, 95% CI 2-sided [-29.57 to 3.31]
Statistical Analysis 8: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 8]; Test type: Superiority or Other; Percent Difference = 8.09, 95% CI 2-sided [-0.52 to 17.81]
Statistical Analysis 9: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 9]; Test type: Superiority or Other; Percent Difference = -7.38, 95% CI 2-sided [-22.86 to 8.29]
Statistical Analysis 10: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 10]; Test type: Superiority or Other; Percent Difference = 0.51, 95% CI 2-sided [-8.82 to 10.08]
Statistical Analysis 11: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 11]; Test type: Superiority or Other; Percent Difference = -20.19, 95% CI 2-sided [-35.45 to -3.95]
Statistical Analysis 12: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 12]; Test type: Superiority or Other; Percent Difference = 5.25, 95% CI 2-sided [-8.50 to 19.06]
Statistical Analysis 13: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 13]; Test type: Superiority or Other; Percent Difference = -3.14, 95% CI 2-sided [-17.51 to 11.13]

36. Secondary Outcome: Percentage of Participants With OPA Titer >= Lower Limit of Quantitation (LLOQ) 1 Month After Toddler Dose
Description: as for outcome 34
Time Frame: 1 Month After Toddler Dose
Population: Evaluable Toddler Immunogenicity Population. Here 'n' signifies participants with a determinate OPA titer to the given serotype during specified follow-up period for each arm, respectively.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Number analyzed (Participants) | 88 | 88
percentage of participants
  4 (n= 67, 61) | 100.00 [94.64 to 100.00] | 100.00 [94.13 to 100.00]
  6B (n= 64, 61) | 98.44 [91.60 to 99.96] | 98.36 [91.20 to 99.96]
  9V (n= 60, 58) | 95.00 [86.08 to 98.96] | 96.55 [88.09 to 99.58]
  14 (n= 62, 62) | 100.00 [94.22 to 100.00] | 100.00 [94.22 to 100.00]
  18C (n= 62, 63) | 98.39 [91.34 to 99.96] | 100.00 [94.31 to 100.00]
  19F (n= 61, 62) | 88.52 [77.78 to 95.26] | 95.16 [86.50 to 98.99]
  23F (n= 65, 63) | 98.46 [91.72 to 99.96] | 98.41 [91.47 to 99.96]
  1 (n= 80, 83) | 87.50 [78.21 to 93.84] | 93.98 [86.50 to 98.02]
  3 (n=78, 79) | 100.00 [95.38 to 100.00] | 98.73 [93.15 to 99.97]
  5 (n= 80, 83) | 96.25 [89.43 to 99.22] | 97.59 [91.57 to 99.71]
  6A (n=78, 74) | 100.00 [95.38 to 100.00] | 100.00 [95.14 to 100.00]
  7F (n= 81, 82) | 100.00 [95.55 to 100.00] | 100.00 [95.60 to 100.00]
  19A (n= 81, 82) | 100.00 [95.55 to 100.00] | 100.00 [95.60 to 100.00]
Statistical Analysis 1: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 1]; Test type: Superiority or Other; Percent Difference = 0.00, 95% CI 2-sided [-5.59 to 5.89]
Statistical Analysis 2: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 2]; Test type: Superiority or Other; Percent Difference = 0.08, 95% CI 2-sided [-6.81 to 7.37]
Statistical Analysis 3: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 3]; Test type: Superiority or Other; Percent Difference = -1.55, 95% CI 2-sided [-10.87 to 7.44]
Statistical Analysis 4: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 4]; Test type: Superiority or Other; Percent Difference = 0.00, 95% CI 2-sided [-5.94 to 5.94]
Statistical Analysis 5: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 5]; Test type: Superiority or Other; Percent Difference = -1.61, 95% CI 2-sided [-8.66 to 4.25]
Statistical Analysis 6: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 6]; Test type: Superiority or Other; Percent Difference = -6.64, 95% CI 2-sided [-17.93 to 3.56]
Statistical Analysis 7: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 7]; Test type: Superiority or Other; Percent Difference = 0.05, 95% CI 2-sided [-6.74 to 7.04]
Statistical Analysis 8: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 1: CI Parameter was percent difference between the groups. Exact 2-sided, 95% CI was computed based on the procedure of Chan and Zhang using the standardized test statistics and gamma=0.000001; Test type: Superiority or Other; Percent Difference = -6.48, 95% CI 2-sided [-16.37 to 2.75]
Statistical Analysis 9: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); Serotype 3: CI Parameter was percent difference between the groups. Exact 2-sided, 95% CI was computed based on the procedure of Chan and Zhang using the standardized test statistics and gamma=0.000001; Test type: Superiority or Other; Percent Difference = 1.27, 95% CI 2-sided [-3.37 to 6.85]
Statistical Analysis 10: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 10]; Test type: Superiority or Other; Percent Difference = -1.34, 95% CI 2-sided [-8.36 to 5.14]
Statistical Analysis 11: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 11]; Test type: Superiority or Other; Percent Difference = 0.00, 95% CI 2-sided [-4.73 to 5.04]
Statistical Analysis 12: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 12]; Test type: Superiority or Other; Percent Difference = 0.00, 95% CI 2-sided [-4.48 to 4.55]
Statistical Analysis 13: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 13]; Test type: Superiority or Other; Percent Difference = 0.00, 95% CI 2-sided [-4.48 to 4.55]

37. Secondary Outcome: Percentage of Participants With OPA Titer >= Lower Limit of Quantitation (LLOQ) 1 Year After Toddler Dose
Description: as for outcome 34
Time Frame: 1 Year After Toddler Dose
Population: as for outcome 32
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Number analyzed (Participants) | 80 | 80
percentage of participants
  4 (n= 66, 59) | 34.8 [23.5 to 47.6] | 42.4 [29.6 to 55.9]
  6B (n= 65, 59) | 41.5 [29.4 to 54.4] | 47.5 [34.3 to 60.9]
  9V (n= 61, 63) | 62.3 [49.0 to 74.4] | 73.0 [60.3 to 83.4]
  14 (n= 59, 54) | 86.4 [75.0 to 94.0] | 90.7 [79.7 to 96.9]
  18C (n= 62, 60) | 38.7 [26.6 to 51.9] | 61.7 [48.2 to 73.9]
  19F (n= 67, 57) | 17.9 [9.6 to 29.2] | 29.8 [18.4 to 43.4]
  23F (n= 67, 62) | 49.3 [36.8 to 61.8] | 77.4 [65.0 to 87.1]
  1 (n= 76, 74) | 10.5 [4.7 to 19.7] | 10.8 [4.8 to 20.2]
  3 (n=76, 70) | 47.4 [35.8 to 59.2] | 48.6 [36.4 to 60.8]
  5 (n= 72, 70) | 20.8 [12.2 to 32.0] | 31.4 [20.9 to 43.6]
  6A (n=70, 70) | 62.9 [50.5 to 74.1] | 81.4 [70.3 to 89.7]
  7F (n= 71, 71) | 93.0 [84.3 to 97.7] | 90.1 [80.7 to 95.9]
  19A (n= 74, 73) | 54.1 [42.1 to 65.7] | 72.6 [60.9 to 82.4]
Statistical Analysis 1: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 1]; Test type: Superiority or Other; Percent Difference = -7.5, 95% CI 2-sided [-24.5 to 9.9]
Statistical Analysis 2: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 2]; Test type: Superiority or Other; Percent Difference = -5.9, 95% CI 2-sided [-23.6 to 11.8]
Statistical Analysis 3: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 3]; Test type: Superiority or Other; Percent Difference = -10.7, 95% CI 2-sided [-27.6 to 6.0]
Statistical Analysis 4: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 4]; Test type: Superiority or Other; Percent Difference = -4.3, 95% CI 2-sided [-17.0 to 8.4]
Statistical Analysis 5: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 5]; Test type: Superiority or Other; Percent Difference = -23.0, 95% CI 2-sided [-40.0 to -4.9]
Statistical Analysis 6: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 6]; Test type: Superiority or Other; Percent Difference = -11.9, 95% CI 2-sided [-27.4 to 3.4]
Statistical Analysis 7: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 7]; Test type: Superiority or Other; Percent Difference = -28.2, 95% CI 2-sided [-43.9 to -11.0]
Statistical Analysis 8: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 8]; Test type: Superiority or Other; Percent Difference = -0.3, 95% CI 2-sided [-10.9 to 10.3]
Statistical Analysis 9: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 9]; Test type: Superiority or Other; Percent Difference = -1.2, 95% CI 2-sided [-17.5 to 15.1]
Statistical Analysis 10: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 10]; Test type: Superiority or Other; Percent Difference = -10.6, 95% CI 2-sided [-25.3 to 4.5]
Statistical Analysis 11: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 11]; Test type: Superiority or Other; Percent Difference = -18.6, 95% CI 2-sided [-33.3 to -3.0]
Statistical Analysis 12: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 12]; Test type: Superiority or Other; Percent Difference = 2.8, 95% CI 2-sided [-7.1 to 13.1]
Statistical Analysis 13: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 13]; Test type: Superiority or Other; Percent Difference = -18.5, 95% CI 2-sided [-33.7 to -2.8]

38. Secondary Outcome: Percentage of Participants With OPA Titer >= Lower Limit of Quantitation (LLOQ) 2 Years After Toddler Dose
Description: as for outcome 34
Time Frame: 2 Years After Toddler Dose
Population: as for outcome 32
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC Group 1 (Preterm Infant) | 13vPnC Group 2 (Term Infant)
Number analyzed (Participants) | 71 | 71
percentage of participants
  4 (n= 46, 54) | 21.7 [10.9 to 36.4] | 29.6 [18.0 to 43.6]
  6B (n= 56, 48) | 35.7 [23.4 to 49.6] | 35.4 [22.2 to 50.5]
  9V (n= 50, 55) | 60.0 [45.2 to 73.6] | 52.7 [38.8 to 66.3]
  14 (n= 49, 45) | 81.6 [68.0 to 91.2] | 84.4 [70.5 to 93.5]
  18C (n= 56, 56) | 21.4 [11.6 to 34.4] | 39.3 [26.5 to 53.2]
  19F (n= 60, 58) | 25.0 [14.7 to 37.9] | 29.3 [18.1 to 42.7]
  23F (n= 58, 59) | 53.4 [39.9 to 66.7] | 74.6 [61.6 to 85.0]
  1 (n= 70, 68) | 8.6 [3.2 to 17.7] | 2.9 [0.4 to 10.2]
  3 (n=69, 66) | 46.4 [34.3 to 58.8] | 51.5 [38.9 to 64.0]
  5 (n= 68, 69) | 7.4 [2.4 to 16.3] | 21.7 [12.7 to 33.3]
  6A (n=68, 62) | 44.1 [32.1 to 56.7] | 64.5 [51.3 to 76.3]
  7F (n= 64, 65) | 68.8 [55.9 to 79.8] | 80.0 [68.2 to 88.9]
  19A (n= 68, 67) | 45.6 [33.5 to 58.1] | 67.2 [54.6 to 78.2]
Statistical Analysis 1: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 1]; Test type: Superiority or Other; Percent Difference = -7.9, 95% CI 2-sided [-25.2 to 9.9]
Statistical Analysis 2: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 2]; Test type: Superiority or Other; Percent Difference = 0.3, 95% CI 2-sided [-18.5 to 19.0]
Statistical Analysis 3: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 3]; Test type: Superiority or Other; Percent Difference = 7.3, 95% CI 2-sided [-12.0 to 26.2]
Statistical Analysis 4: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 4]; Test type: Superiority or Other; Percent Difference = -2.8, 95% CI 2-sided [-19.1 to 13.3]
Statistical Analysis 5: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 5]; Test type: Superiority or Other; Percent Difference = -17.9, 95% CI 2-sided [-34.6 to -0.3]
Statistical Analysis 6: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 6]; Test type: Superiority or Other; Percent Difference = -4.3, 95% CI 2-sided [-20.6 to 12.1]
Statistical Analysis 7: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 7]; Test type: Superiority or Other; Percent Difference = -21.1, 95% CI 2-sided [-37.8 to -3.2]
Statistical Analysis 8: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 8]; Test type: Superiority or Other; Percent Difference = 5.6, 95% CI 2-sided [-2.7 to 15.2]
Statistical Analysis 9: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 9]; Test type: Superiority or Other; Percent Difference = -5.1, 95% CI 2-sided [-22.0 to 12.0]
Statistical Analysis 10: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 10]; Test type: Superiority or Other; Percent Difference = -14.4, 95% CI 2-sided [-26.7 to -2.4]
Statistical Analysis 11: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 11]; Test type: Superiority or Other; Percent Difference = -20.4, 95% CI 2-sided [-36.8 to -3.0]
Statistical Analysis 12: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 12]; Test type: Superiority or Other; Percent Difference = -11.3, 95% CI 2-sided [-26.4 to 4.1]
Statistical Analysis 13: Comparison: 13vPnC Group 1 (Preterm Infant) vs 13vPnC Group 2 (Term Infant); [analysis description as in outcome 34, analysis 13]; Test type: Superiority or Other; Percent difference = -21.6, 95% CI 2-sided [-37.7 to -4.6]

ADVERSE EVENTS:
Time Frame: AEs/SAEs: recorded from 13vPnC infant dose 1 to 2-year follow-up after toddler dose. Participants recorded pre-specified AEs in electronic diary: local reactions; systemic events (up to 7 days after each vaccine dose)
Description: SAEs and AEs were grouped by system organ class and summarized. AEs included AEs collected in electronic diary (local,systemic reactions for 13vPnC; systematic assessment) and AEs collected on case report form at each visit (nonsystematic assessment). Participants who received specified dose and had safety data available were evaluable for safety.
Groups:
- 13vPnC Group 1 (Preterm Infant) - Infant Series: Preterm infant participants (GA <37 weeks) who received single 0.5 mL dose of 13vPnC intramuscularly at 2, 3 and 4 months of age (infant series), assessed from Infant Dose 1 through the blood draw 1 month after Infant Dose 3.
- 13vPnC Group 2 (Term Infant) - Infant Series: Term infant participants (GA >=37 weeks) who received single 0.5 mL dose of 13vPnC intramuscularly at 2, 3, 4 months of age (infant series), assessed from Infant Dose 1 through the blood draw 1 month after Infant Dose 3.
- 13vPnC Group 1 (Preterm Infant) - After Infant Series: Preterm infant participants (GA <37 weeks) who received single 0.5 mL dose of 13vPnC intramuscularly at 2, 3 and 4 months of age (infant series), assessed from blood draw 1 month after infant Dose 3 to before toddler dose.
- 13vPnC Group 2 (Term Infant) - After Infant Series: Term infant participants (GA >=37 weeks) who received single 0.5 mL dose of 13vPnC intramuscularly at 2, 3, 4 months of age (infant series), assessed from blood draw 1 month after infant Dose 3 to before toddler dose.
- 13vPnC Group 1 (Preterm Infant) - Toddler Dose: Preterm infant participants (GA <37 weeks) who received single 0.5 mL dose of 13vPnC intramuscularly at 2, 3, 4 months of age (infant series) and 12 months of age (toddler dose), assessed from the toddler dose through the blood draw 1 month after toddler dose.
- 13vPnC Group 2 (Term Infant) - Toddler Dose: Term infant participants (GA >=37 weeks) who received single 0.5 mL dose of 13vPnC intramuscularly at 2, 3, 4 months of age (infant series) and 12 months of age (toddler dose), assessed from the toddler dose through the blood draw 1 month after toddler dose.
- 13vPnC Group 1 (Preterm Infant) - 1 Year Follow-up: Preterm infant participants (GA <37 weeks) who received single 0.5 mL dose of 13vPnC intramuscularly at 2, 3, 4 months of age (infant series) and 12 months of age (toddler dose), assessed from blood draw 1 month after the toddler dose to 1-year follow-up.
- 13vPnC Group 2 (Term Infant) - 1 Year Follow-up: Term infant participants (GA >=37 weeks) who received single 0.5 mL dose of 13vPnC intramuscularly at 2, 3, 4 months of age (infant series) and 12 months of age (toddler dose), assessed from blood draw 1 month after the toddler dose to 1-year follow-up.
- 13vPnC Group 1 (Preterm Infant) - 2 Year Follow-up: Preterm infant participants (GA <37 weeks) who received single 0.5 mL dose of 13vPnC intramuscularly at 2, 3, 4 months of age (infant series) and 12 months of age (toddler dose), assessed from 1-year follow-up after toddler dose to 2-year follow-up after toddler dose.
- 13vPnC Group 2 (Term Infant) - 2 Year Follow-up: Term infant participants (GA >=37 weeks) who received single 0.5 mL dose of 13vPnC intramuscularly at 2, 3, 4 months of age (infant series) and 12 months of age (toddler dose), assessed from 1-year follow-up after toddler dose to 2-year follow-up after toddler dose.
Arm/Group | 13vPnC Group 1 (Preterm Infant) - Infant Series | 13vPnC Group 2 (Term Infant) - Infant Series | 13vPnC Group 1 (Preterm Infant) - After Infant Series | 13vPnC Group 2 (Term Infant) - After Infant Series | 13vPnC Group 1 (Preterm Infant) - Toddler Dose | 13vPnC Group 2 (Term Infant) - Toddler Dose | 13vPnC Group 1 (Preterm Infant) - 1 Year Follow-up | 13vPnC Group 2 (Term Infant) - 1 Year Follow-up | 13vPnC Group 1 (Preterm Infant) - 2 Year Follow-up | 13vPnC Group 2 (Term Infant) - 2 Year Follow-up
Serious Adverse Events (participants affected / at risk) | 14/100 | 5/100 | 8/100 | 9/100 | 2/99 | 1/97 | 13/99 | 8/97 | 6/88 | 8/88
Other Adverse Events (participants affected / at risk) | 98/100 | 99/100 | 13/100 | 11/100 | 93/99 | 92/97 | 2/99 | 0/97 | 1/88 | 1/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC Group 1 (Preterm Infant) - Infant Series (N=100) | 13vPnC Group 2 (Term Infant) - Infant Series (N=100) | 13vPnC Group 1 (Preterm Infant) - After Infant Series (N=100) | 13vPnC Group 2 (Term Infant) - After Infant Series (N=100) | 13vPnC Group 1 (Preterm Infant) - Toddler Dose (N=99) | 13vPnC Group 2 (Term Infant) - Toddler Dose (N=97) | 13vPnC Group 1 (Preterm Infant) - 1 Year Follow-up (N=99) | 13vPnC Group 2 (Term Infant) - 1 Year Follow-up (N=97) | 13vPnC Group 1 (Preterm Infant) - 2 Year Follow-up (N=88) | 13vPnC Group 2 (Term Infant) - 2 Year Follow-up (N=88)
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Intussusception (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Adenoviral upper respiratory infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 4 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 3 | 0 | 0 | 0 | 4 | 0 | 0 | 2
Pneumonia respiratory syncytial viral (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 1
Human herpesvirus 6 infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Viral rash (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia mycoplasmal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Encephalitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Meningitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian cyst torsion (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hip dysplasia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral palsy (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Autism spectrum disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
CSF shunt operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC Group 1 (Preterm Infant) - Infant Series (N=100) | 13vPnC Group 2 (Term Infant) - Infant Series (N=100) | 13vPnC Group 1 (Preterm Infant) - After Infant Series (N=100) | 13vPnC Group 2 (Term Infant) - After Infant Series (N=100) | 13vPnC Group 1 (Preterm Infant) - Toddler Dose (N=99) | 13vPnC Group 2 (Term Infant) - Toddler Dose (N=97) | 13vPnC Group 1 (Preterm Infant) - 1 Year Follow-up (N=99) | 13vPnC Group 2 (Term Infant) - 1 Year Follow-up (N=97) | 13vPnC Group 1 (Preterm Infant) - 2 Year Follow-up (N=88) | 13vPnC Group 2 (Term Infant) - 2 Year Follow-up (N=88)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Craniotabes (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye discharge (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 1 | 1 | 2 | 2 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infantile colic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Irritability (General disorders) | 5 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 4 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Food allergy (Immune system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Milk allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 7 | 6 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 5 | 1 | 0 | 3 | 3 | 2 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Exanthema subitum (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 6 | 1 | 0 | 3 | 2 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 6 | 5 | 0 | 2 | 6 | 4 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 1 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 8 | 9 | 4 | 0 | 3 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 5 | 4 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 8 | 10 | 1 | 0 | 5 | 4 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Viral rash (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotonia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subdural hygroma (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Beckwith-Wiedemann syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Teething (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Herpangina (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Developmental delay (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Tenderness- Any (Skin and subcutaneous tissue disorders) | 46/94 | 37/88 | 0/0 | 0/0 | 60/86 | 47/85 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 1 Infant Series and Toddler Dose
Tenderness- Any (Skin and subcutaneous tissue disorders) | 41/85 | 34/88 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Tenderness- Any (Skin and subcutaneous tissue disorders) | 32/82 | 24/84 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 3 Infant Series
Tenderness- Mild (Skin and subcutaneous tissue disorders) | 43/93 | 28/88 | 0/0 | 0/0 | 57/86 | 44/85 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 1 Infant Series and Toddler Dose
Tenderness- Mild (Skin and subcutaneous tissue disorders) | 37/85 | 26/84 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Tenderness- Mild (Skin and subcutaneous tissue disorders) | 29/81 | 22/84 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 3 Infant Series
Tenderness- Moderate (Skin and subcutaneous tissue disorders) | 16/90 | 14/85 | 0/0 | 0/0 | 16/77 | 8/70 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 1 Infant Series and Toddler Dose
Tenderness- Moderate (Skin and subcutaneous tissue disorders) | 11/77 | 13/83 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Tenderness- Moderate (Skin and subcutaneous tissue disorders) | 7/75 | 4/78 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 3 Infant Series
Tenderness- Severe (Skin and subcutaneous tissue disorders) | 0/86 | 0/85 | 0/0 | 0/0 | 2/74 | 0/69 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 1 Infant Series and Toddler Dose
Tenderness- Severe (Skin and subcutaneous tissue disorders) | 0/73 | 1/77 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Tenderness- Severe (Skin and subcutaneous tissue disorders) | 0/73 | 0/77 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 3 Infant Series
Swelling- Any (Skin and subcutaneous tissue disorders) | 37/94 | 26/89 | 0/0 | 0/0 | 35/81 | 28/80 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 1 Infant Series and Toddler Dose
Swelling- Any (Skin and subcutaneous tissue disorders) | 30/84 | 35/82 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Swelling- Any (Skin and subcutaneous tissue disorders) | 25/83 | 35/85 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 3 Infant Series
Swelling- Mild (Skin and subcutaneous tissue disorders) | 34/91 | 25/89 | 0/0 | 0/0 | 31/80 | 26/79 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 1 Infant Series and Toddler Dose
Swelling- Mild (Skin and subcutaneous tissue disorders) | 28/83 | 35/82 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0/0 — Dose 2 Infant Series
Swelling- Mild (Skin and subcutaneous tissue disorders) | 22/82 | 35/85 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 3 Infant Series
Swelling- Moderate (Skin and subcutaneous tissue disorders) | 8/91 | 7/85 | 0/0 | 0/0 | 10/76 | 7/74 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 1 Infant Series and Toddler Dose
Swelling- Moderate (Skin and subcutaneous tissue disorders) | 6/75 | 2/76 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Swelling- Moderate (Skin and subcutaneous tissue disorders) | 4/75 | 4/79 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 3 Infant Series
Swelling- Severe (Skin and subcutaneous tissue disorders) | 0/86 | 0/85 | 0/0 | 0/0 | 1/74 | 0/69 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 1 Infant Series and Toddler Dose
Swelling- Severe (Skin and subcutaneous tissue disorders) | 0/73 | 0/76 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Swelling- Severe (Skin and subcutaneous tissue disorders) | 0/73 | 0/77 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 3 Infant Series
Redness- Any (Skin and subcutaneous tissue disorders) | 31/92 | 26/87 | 0/0 | 0/0 | 44/85 | 41/83 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 1 Infant Series and Toddler Dose
Redness- Any (Skin and subcutaneous tissue disorders) | 23/82 | 33/82 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Redness- Any (Skin and subcutaneous tissue disorders) | 27/82 | 40/87 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 3 Infant Series
Redness- Mild (Skin and subcutaneous tissue disorders) | 29/90 | 25/87 | 0/0 | 0/0 | 44/85 | 40/83 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 1 Infant Series and Toddler Dose
Redness- Mild (Skin and subcutaneous tissue disorders) | 23/82 | 31/82 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Redness- Mild (Skin and subcutaneous tissue disorders) | 27/82 | 40/87 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 3 Infant Series
Redness- Moderate (Skin and subcutaneous tissue disorders) | 3/88 | 4/85 | 0/0 | 0/0 | 5/75 | 8/75 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 1 Infant Series and Toddler Dose
Redness- Moderate (Skin and subcutaneous tissue disorders) | 2/73 | 2/76 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Redness- Moderate (Skin and subcutaneous tissue disorders) | 1/74 | 3/79 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 3 Infant Series
Redness- Severe (Skin and subcutaneous tissue disorders) | 0/86 | 0/85 | 0/0 | 0/0 | 0/74 | 0/69 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 1 Infant Series and Toddler Dose
Redness- Severe (Skin and subcutaneous tissue disorders) | 0/73 | 0/76 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Redness- Severe (Skin and subcutaneous tissue disorders) | 0/73 | 0/77 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 3 Infant Series
Fever >=38 degrees C (General disorders) | 10/86 | 12/88 | 0/0 | 0/0 | 23/80 | 34/78 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 1 Infant Series and Toddler Dose
Fever >=38 degrees C (General disorders) | 22/79 | 25/79 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Fever >=38 degrees C (General disorders) | 22/79 | 25/81 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 3 Infant Series
Fever >=38 degrees C, =<39 degrees C (General disorders) | 9/86 | 12/88 | 0/0 | 0/0 | 22/80 | 33/77 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 1 Infant Series and Toddler Dose
Fever >=38 degrees C, =<39 degrees C (General disorders) | 22/79 | 24/79 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Fever >=38 degrees C, =<39 degrees C (General disorders) | 21/78 | 25/81 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 3 Infant Series
Fever >=39 degrees C, =<40 degrees C (General disorders) | 1/86 | 0/85 | 0/0 | 0/0 | 1/74 | 3/71 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 1 Infant Series and Toddler Dose
Fever >=39 degrees C, =<40 degrees C (General disorders) | 0/73 | 1/76 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Fever >=39 degrees C, =<40 degrees C (General disorders) | 1/75 | 2/78 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 3 Infant Series
Fever >40 degrees C (General disorders) | 0/86 | 0/85 | 0/0 | 0/0 | 0/74 | 1/70 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 1 Infant Series and Toddler Dose
Fever >40 degrees C (General disorders) | 0/73 | 0/76 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Fever >40 degrees C (General disorders) | 0/74 | 0/77 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 — Dose 3 Infant Series
Decreased Appetite- Any (General disorders) | 56/92 | 37/89 | 0/0 | 0/0 | 50/87 | 52/86 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 1 Infant Series and Toddler Dose
Decreased Appetite- Any (General disorders) | 55/89 | 39/84 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Decreased Appetite- Any (General disorders) | 40/82 | 40/84 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 3 Infant Series
Decreased Appetite- Mild (General disorders) | 50/91 | 31/88 | 0/0 | 0/0 | 43/86 | 47/84 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 1 Infant Series and Toddler Dose
Decreased Appetite- Mild (General disorders) | 49/88 | 35/84 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Decreased Appetite- Mild (General disorders) | 30/82 | 39/84 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 3 Infant Series
Decreased Appetite- Moderate (General disorders) | 18/88 | 15/87 | 0/0 | 0/0 | 20/78 | 17/73 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 1 Infant Series and Toddler Dose
Decreased Appetite- Moderate (General disorders) | 20/79 | 15/78 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Decreased Appetite- Moderate (General disorders) | 13/74 | 13/79 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 3 Infant Series
Decreased Appetite- Severe (General disorders) | 1/86 | 0/85 | 0/0 | 0/0 | 1/75 | 1/69 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 1 Infant Series and Toddler Dose
Decreased Appetite- Severe (General disorders) | 1/73 | 0/76 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Decreased Appetite- Severe (General disorders) | 1/74 | 1/77 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 3 Infant Series
Increased Sleep- Any (General disorders) | 65/96 | 66/95 | 0/0 | 0/0 | 48/83 | 56/86 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 1 Infant Series and Toddler Dose
Increased Sleep- Any (General disorders) | 63/85 | 57/89 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Increased Sleep- Any (General disorders) | 46/88 | 51/88 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 3 Infant Series
Increased Sleep- Mild (General disorders) | 58/96 | 57/93 | 0/0 | 0/0 | 44/82 | 50/84 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 1 Infant Series and Toddler Dose
Increased Sleep- Mild (General disorders) | 58/83 | 52/88 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Increased Sleep- Mild (General disorders) | 43/88 | 45/87 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 3 Infant Series
Increased Sleep- Moderate (General disorders) | 26/87 | 27/88 | 0/0 | 0/0 | 14/76 | 18/74 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 1 Infant Series and Toddler Dose
Increased Sleep- Moderate (General disorders) | 27/78 | 23/78 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Increased Sleep- Moderate (General disorders) | 13/77 | 16/80 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 3 Infant Series
Increased Sleep- Severe (General disorders) | 2/86 | 2/85 | 0/0 | 0/0 | 0/74 | 2/70 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 1 Infant Series and Toddler Dose
Increased Sleep- Severe (General disorders) | 2/73 | 1/76 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Increased Sleep- Severe (General disorders) | 1/73 | 1/77 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 3 Infant Series
Irritability or Decreased Sleep- Any (General disorders) | 80/95 | 80/97 | 0/0 | 0/0 | 76/90 | 73/91 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 1 Infant Series and Toddler Dose
Irritability or Decreased Sleep- Any (General disorders) | 85/95 | 74/95 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Irritability or Decreased Sleep- Any (General disorders) | 73/92 | 77/95 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 3 Infant Series
Irritability or Decreased Sleep- Mild (General disorders) | 72/93 | 66/95 | 0/0 | 0/0 | 67/90 | 68/89 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 1 Infant Series and Toddler Dose
Irritability or Decreased Sleep- Mild (General disorders) | 73/90 | 66/92 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Irritability or Decreased Sleep- Mild (General disorders) | 65/90 | 68/91 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 3 Infant Series
Irritability or Decreased Sleep-Moderate (General disorders) | 40/92 | 43/91 | 0/0 | 0/0 | 35/78 | 36/80 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 1 Infant Series and Toddler Dose
Irritability or Decreased Sleep-Moderate (General disorders) | 55/85 | 38/86 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Irritability or Decreased Sleep-Moderate (General disorders) | 27/80 | 31/87 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 3 Infant Series
Irritability or Decreased Sleep- Severe (General disorders) | 7/86 | 5/85 | 0/0 | 0/0 | 5/76 | 3/69 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 1 Infant Series and Toddler Dose
Irritability or Decreased Sleep- Severe (General disorders) | 13/74 | 2/76 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Irritability or Decreased Sleep- Severe (General disorders) | 5/74 | 5/78 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 3 Infant Series
Use of Antipyretic Medication (General disorders) | 22/90 | 22/90 | 0/0 | 0/0 | 40/82 | 40/79 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 1 Infant Series and Toddler Dose
Use of Antipyretic Medication (General disorders) | 41/84 | 38/83 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 2 Infant Series
Use of Antipyretic Medication (General disorders) | 34/84 | 31/81 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Dose 3 Infant Series

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.